#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for a Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Mepolizumab Administered Subcutaneously in Subjects with Moderate to Severe Atopic Dermatitis

Compound Number : SB240563

Effective Date : 28-FEB-2018

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and outputs to be included in the Clinical Study Report for Protocol GSK Document Number 2015N268158\_02
- This RAP is intended to describe the efficacy, safety and tolerability, pharmacokinetic and pharmacodynamic analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **RAP Author(s):**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | | |
| Associate Statistician (Immuno Inflammation,<br>Quantitative Sciences India) | NA | NA |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

# **RAP Team Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Clinical Investigation Leader (Immuno Inflammation, Immuno Immunology) | 22-FEB-2018 | eTMF |
| Project Physician Leader (Clinical Pharmacology<br>Modelling and Simulation) | 28-FEB-2018 | E-Mail |
| SERM Director (CMO GCSP) | 26-FEB-2018 | eTMF |
| Operational Scientist Leader (PCPS) | 22-FEB-2018 | eTMF |
| Data Quality Leader (Immuno Inflammation and Dermatology, Data Management) | 28-FEB-2018 | eTMF |
| Pharmacokinetist (Clinical Pharmacology<br>Modelling and Simulation) | 24-FEB-2018 | eTMF |
| Lead Programmer (Future Pipeline Discovery,<br>Quantitative Sciences India) | 28-FEB-2018 | eTMF |

# **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval Method |
|---|---|---|
| Statistical Leader (Immuno Inflammation,<br>Quantitative Sciences India) | 25-FEB-2018 | eTMF |
| Biostatistics and Programming Manager (Future Pipeline Discovery, Quantitative Sciences India) | 23-FEB-2018 | eTMF |

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DDUCTIO | DN | 6 |
| 2. | SUMN | MARY OF | KEY PROTOCOL INFORMATION | 6 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | ۷.۷. | 2.2.1. | | |
| | | 2.2.1. | Final Reporting Objectives & Endpoints Following Study | |
| | | ۷.۷.۷. | Termination | Q |
| | 2.3. | Study F | Design | |
| | 2.4. | | cal Hypotheses / Statistical Analyses | |
| | 2.4. | Statistic | Lai Hypotheses / Statistical Arialyses | 12 |
| 3. | PLAN | NED AN | ALYSES | 12 |
| | 3.1. | Interim | Analyses | 12 |
| | 3.2. | Final Ar | nalyses | 14 |
| 4. | | | PULATIONS | |
| | 4.1. | Protoco | ol Deviations | 15 |
| 5. | CONS | IDEDAT | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| J. | | | IS | 15 |
| | 5.1. | | reatment & Sub-group Display Descriptors | |
| | 5.2. | | e Definitions | |
| | J.Z. | 5.2.1. | | |
| | 5.3. | - | Considerations for Data Analyses and Data Handling | 10 |
| | 0.0. | | ntions | 16 |
| 6. | STUD | Y POPU | LATION ANALYSES | 17 |
| | 6.1. | Overvie | ew of Planned Study Population Analyses | 17 |
| 7 | FFFIC | | ALVOCO | 47 |
| 7. | | | ALYSES | |
| | 7.1. | - | / Efficacy Analyses | |
| | | 7.1.1. | | |
| | | 7.1.2. | <b>,</b> | |
| | | 7.1.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.1.4. | Population of Interest | |
| | | 7.1.5. | Statistical Analyses / Methods | |
| | 7.2. | Sacand | 7.1.5.1. Statistical Methodology Specification | |
| | 1.2. | 7.2.1. | lary Efficacy Analyses<br>Endpoint / Variables | |
| | | 7.2.1.<br>7.2.2. | Summary Measure | |
| | | 7.2.2.<br>7.2.3. | Strategy for Intercurrent (Post-Randomization) Events | |
| | | 7.2.3.<br>7.2.4. | Population of Interest | |
| | | 7.2.5. | Statistical Analyses / Methods | |
| | | 1.2.0. | 7.2.5.1. Statistical Methodology Specification | |
| | 7.3. | Explora | tory Efficacy Analyses | |
| | | 7.3.1. | Endpoint / Variables | |
| | | 7.3.2. | Summary Measure | |
| | | 7.3.3. | Strategy for Intercurrent (Post-Randomization) Events | |

#### CONFIDENTIAL

| | | 7.3.4. | Population | of Interest | .20 |
|---|---|---|---|---|---|
| | | | 7.3.4.1. | Statistical Analyses / Methods | .20 |
| | | | 7.3.4.2. | Statistical Methodology Specification | .20 |
| _ | | | | | |
| 8. | | | | | |
| | 8.1. | | | alyses | |
| | 8.2. | | | Special Interest Analyses | |
| | 8.3. | | | Analyses | |
| | 8.4. | Other Sa | fety Analys | es | .21 |
| | | 8.4.1. | ECG | | .21 |
| | 8.5. | Immunog | genicity Ana | alyses | .22 |
| 9. | DHARI | MACOKIN | IETIC ANA | LYSES | 23 |
| J. | 9.1. | | | cokinetic Analyses | |
| | J. 1. | 9.1.1. | • | Variables | |
| | | 9.1.1. | 9.1.1.1. | Drug Concentration Measures | |
| | | | 9.1.1.1. | Derived Pharmacokinetic Parameters | |
| | | 0.4.0 | O | | |
| | | 9.1.2. | | Measure | |
| | | 9.1.3. | | of Interest | |
| | | 9.1.4. | | or Intercurrent (Post-Randomization) Events | |
| | | 9.1.5. | Statistical | Analyses / Methods | .23 |
| 10. | PHARI | MACODY | NAMIC AN | D BIOMARKER ANALYSES | .24 |
| | 10.1. | Explorate | ory Pharma | codynamic and Biomarker Analyses | .24 |
| | | 10.1.1. | | Variables | |
| | | 10.1.2. | | Measure | |
| | | 10.1.3. | • | of Interest | |
| | | 10.1.4. | • | Analyses / Methods | |
| | | . • | | Statistical Methodology Specification | |
| 44 | DEEE | DENOCE | | | 200 |
| 11. | KEFE | KENCES. | | | . 26 |
| 12. | APPE | NDICES | | | 27 |
| | 12.1. | | | lle of Activities | |
| | 12.2. | | | ment Windows | |
| | | | | of Assessment Windows for Analyses | |
| | 12.3. | | | Phases and Treatment Emergent Adverse | |
| | | Events | | <u> </u> | .32 |
| | | 12.3.1. | Study Pha | ses | .32 |
| | | | | Study Phases for Efficacy Assessments | |
| | | 12.3.2. | | Emergent Flag for Adverse Events | |
| | 12.4. | _ | | splay Standards & Handling Conventions | |
| | | 12.4.1. | | Process | |
| | | 12.4.2. | | Standards | |
| | | 12.4.3. | | Standards for Pharmacokinetic | |
| | 12.5. | | | I and Transformed Data | |
| | 12.0. | 12.5.1. | | rana Transformed Bata | |
| | | 12.5.1. | | ulation | |
| | | 12.5.2. | | uiatioii | |
| | | 12.5.3.<br>12.5.4. | | | |
| | | 12.5.4.<br>12.5.5. | | kinetic | |
| | | 12.5.6. | rnarmaco | dynamic and Biomarker | . J/ |

#### CONFIDENTIAL

| വ | 05 | $\mathbf{a}$ | ·⊏ | r |
|---|----|--------------|----|---|
| | 17 | u | _ | |

| 12.6. | Appendix | c 6: Reporting Standards for Missing Data | .38 |
|--------|----------|-------------------------------------------------|-----|
| | 12.6.1. | Premature Withdrawals | |
| | 12.6.2. | Handling of Missing Data | .38 |
| | | 12.6.2.1. Handling of Missing and Partial Dates | .38 |
| 12.7. | Appendix | 7: Values of Potential Clinical Importance | .39 |
| | 12.7.1. | Laboratory Values | .39 |
| | 12.7.2. | Vital Signs | .39 |
| 12.8. | Appendix | c8: Abbreviations & Trade Marks | .40 |
| | 12.8.1. | Abbreviations | .40 |
| | 12.8.2. | Trademarks | .41 |
| 12.9. | Appendix | र 9: List of Data Displays | .42 |
| | 12.9.1. | Data Display Numbering | .42 |
| | 12.9.2. | Mock Example Shell Referencing | .42 |
| | 12.9.3. | Deliverables | |
| | 12.9.4. | Study Population Tables | .43 |
| | 12.9.5. | Efficacy Tables | .45 |
| | 12.9.6. | Safety Tables | .46 |
| | 12.9.7. | Safety Figures | .51 |
| | 12.9.8. | Pharmacokinetic Tables | .51 |
| | 12.9.9. | Pharmacokinetic Figures | .52 |
| | 12.9.10. | Pharmacodynamic and Biomarker Tables | .52 |
| | 12.9.11. | Pharmacodynamic and Biomarker Figures | .53 |
| | 12.9.12. | ICH Listings | .54 |
| | 12.9.13. | Non-ICH Listings | .57 |
| 12.10. | Appendix | c 10: Example Mock Shells for Data Displays | .59 |

#### 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol:

| Revision Chronology: | |
|---|---|
| 2015N268158_00 2016-AUG-25 | Original |
| 2015N268158_01 | Amendment No. 1 |
| Protocol amendment 1 includes recommendations from the US Food and Drug Administration (FDA) and other clarifications. | |
| 2015N268158_02 2017-JUN-22 Ame | Amendment No. 2 |

- The addition of administrative interim analyses to enable review of subject efficacy and safety data summaries.
- Minor clarifications regarding: collection of ECGs in triplicate for all ECG timepoints; general order
  of study procedures; checks for BSA and EASI eligibility utilizing eCRF auto calculated totals at
  Screening and Baseline visits.
- Increase in anticipated number of subjects screened from approximately 75 subjects to approximately 140 subjects (no change in target number of subjects randomized).
- Reminders inserted into the study schematic and Time and Events tables, indicating no IP dose will be administered at Week 16 and Week 20.
- Removed requirement for subject data entry into the Daily Sign and Symptom
- Severity Diary for at least 7 consecutive days immediately prior to the Baseline visit.

Following a formal interim analysis (10-NOV-2017) after approximately 50% of subjects were randomised and had the opportunity to complete the Week 8 visit, the study met the planned futility stopping criteria and the study was terminated. As a result of the study being terminated, only a sub-set of planned protocol defined objectives and endpoints will be included for the final reporting.

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

Changes from the originally planned statistical analysis specified in the protocol are outlined in Table 1.

Table 1 Changes to Protocol Defined Analysis Plan

| Protocol | Re | porting & Analysis Plan | | |
|---|---|---|---|---|
| Statistical Analysis Pla | | atistical Analysis Plan | Rationale for Cha | nges |
| <ul> <li>Exploratory Objective Proportion of subject have an IGA score of and at least a 2-grade improvement at each visit by baseline blood eosinophil count</li> <li>Exploratory Objective percentage change score compared to oblood eosinophils at</li> </ul> | ves: vts who of 0 or 1 de h study od ves: Mean in EASI change in | These endpoints are not being considered for final reporting | Due to the limi responders, the endpoints will summarised | ted<br>ese |
| Exploratory Objective change in weekly averaged and a second change in weekly averaged and a second change in weekly averaged and second change in the | verage of imeric core f Daily Severity | This endpoint is not considered for final reporting | Mean change<br>for all study vis<br>include Week<br>this is conside<br>scope for final | sit will also<br>16 and hence<br>red as out of |
| Exploratory Objectiv | ves • | Additional Exploratory Objective included: Clinician Global Impression of Change is an exploratory endpoint which is not included while defining the objective/ endpoint | This is collected protocol so incomprehensial reporting | • |
| Section 9.3.1: In all<br>definitions "all subje<br>used | | In all population definition "all<br>subjects" term has been<br>changed to "all participants" | Changed as portion RAP template | |
| Section 9.3.1: Per-P Population definition | | Per-Protocol Population is removed | There is no pla<br>sensitivity ana<br>primary object | lysis for the |
| Section 9.3.1: PK Podefinition | opulation | PK Population definition updated | Changed as part RAP template to take accour miss-dosed part RAP template | definition and<br>it of potential |
| Section 9.1: Mentior Credible Interval for response rate and the difference in respon primary efficacy end later in Section 9.4 r as 80% Credible Interval the response rate and difference in response. | the ne se rate for lpoint and mentions erval for nd the | 80% Credible Interval for the response rate and the difference in response rate is provided for primary efficacy endpoint | There was ince<br>the protocol ar<br>specified as 80<br>Interval for the<br>rate and the di<br>response rate | nd should be<br>0% Credible<br>response |

# 2.2. Study Objective(s) and Endpoint(s)

# 2.2.1. Protocol Defined Objectives and Endpoints

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine the efficacy of<br>mepolizumab SC in subjects with<br>moderate to severe AD | Proportion of subjects who achieve treatment success defined as an Investigator's Global Assessment (IGA) score of 0 or 1 and at least a 2-grade improvement at Week 16. |
| Secondary Objectives | Secondary Endpoints |
| To estimate the efficacy of mepolizumab SC | <ul> <li>Mean percentage change in Eczema Area and Severity Index (EASI) score from baseline to each study visit.</li> <li>Proportion of subjects with an IGA score of 0 or 1 and at least a 2-grade improvement at each study visit.</li> </ul> |
| To describe the safety and tolerability of mepolizumab SC | <ul> <li>Incidence, frequency, and nature of adverse events (AEs) including local injection site reactions and systemic reactions.</li> <li>Change from baseline in laboratory parameters (hematology and chemistry) and frequency of clinically significant abnormal test results.</li> <li>Change from baseline in vital signs and frequency of clinically significant abnormal results.</li> </ul> |
| | Immunogenicity as measured by anti-mepolizumab |
| | antibodies. |
| Exploratory Objectives | Exploratory Endpoints |
| To further estimate the efficacy of mepolizumab SC | <ul> <li>Proportion of subjects with ≥50% improvement in EASI from baseline to each study visit.</li> <li>Proportion of subjects with ≥75% improvement in EASI from baseline to each study visit.</li> <li>Mean change in percent of total body surface area (% BSA) affected from baseline to each study visit.</li> <li>Mean change in weekly average of daily itch/pruritus numeric rating scale [NRS] score (based on Item #1 of Daily Sign and Symptom Severity Diary) from baseline to Week 16.</li> <li>Mean change in weekly average of daily itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary) from baseline to each study visit.</li> </ul> |
| To evaluate disease flare/relapse<br>during and after treatment with<br>mepolizumab SC | <ul> <li>Proportion of subjects who have an IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2-grade improvement during the Treatment and Follow-up Periods.</li> <li>Proportion of subjects who have an increase in EASI score of &gt;=25% from baseline during the Treatment and Follow-up Periods.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To characterize the relationship<br>between efficacy and blood eosinophil<br>count | <ul> <li>Proportion of subjects who have an IGA score of 0 or 1 and at least a 2-grade improvement at each study visit by baseline blood eosinophil count.</li> <li>Mean percentage change in EASI score from baseline to each study visit by baseline blood eosinophil count.</li> <li>Mean percentage change in EASI score compared to change in blood eosinophils at each visit.</li> </ul> |
| To investigate the pharmacokinetics of<br>mepolizumab in subjects with<br>moderate to severe AD | Plasma concentration of mepolizumab |
| To investigate the pharmacodynamics<br>of mepolizumab in the blood and in<br>AD lesional skin biopsies | <ul> <li>Ratio to baseline in blood eosinophil counts</li> <li>IL-5 levels (serum free and total)</li> <li>Levels of circulating biomarkers in the blood including immunoglobulin (IgE), eosinophilic cationic protein (ECP), and levels of chemokines such as thymus and activation-regulated chemokine (TARC)</li> <li>Gene expression biomarkers in skin biopsies</li> </ul> |
| To describe the effect of<br>mepolizumab SC on Patient reported<br>Outcomes (PROs) | <ul> <li>Change over time in Daily Sign and Symptom<br/>Severity Diary</li> <li>Change over time in Patient Global Impression of<br/>Severity and Patient Global Impression of Change</li> </ul> |

# 2.2.2. Final Reporting Objectives & Endpoints Following Study Termination

| Objectives Endpoints | |
|---|---|
| Primary Objectives | Primary Endpoints |
| To determine the efficacy of<br>mepolizumab SC in subjects with<br>moderate to severe AD | <ul> <li>Proportion of subjects who achieve treatment success defined as an Investigator's Global</li> <li>Assessment (IGA) score of 0 or 1 and at least a 2-grade improvement at Week 16.</li> </ul> |
| Secondary Objectives | Secondary Endpoints |
| To estimate the efficacy of mepolizumab SC | <ul> <li>Mean percentage change in Eczema Area and Severity Index (EASI) score from baseline to each study visit.</li> <li>Proportion of subjects with an IGA score of 0 or 1 and at least a 2-grade improvement at each study visit.</li> </ul> |
| To describe the safety and tolerability of mepolizumab SC | <ul> <li>Incidence, frequency, and nature of adverse events (AEs) including local injection site reactions and systemic reactions.</li> <li>Change from baseline in laboratory parameters (hematology and chemistry) and frequency of clinically significant abnormal test results.</li> <li>Change from baseline in vital signs and frequency of clinically significant abnormal results.</li> <li>Immunogenicity as measured by anti-mepolizumab antibodies.</li> </ul> |

| Objectives | Endpoints |
|---|---|
| Exploratory Objectives | Exploratory Endpoints |
| To further estimate the efficacy of mepolizumab SC | <ul> <li>Proportion of subjects with ≥50% improvement in EASI from baseline to each study visit.</li> <li>Proportion of subjects with ≥75% improvement in EASI from baseline to each study visit.</li> <li>Mean change in percent of total body surface area (% BSA) affected from baseline to each study visit.</li> <li>Mean change in weekly average of daily itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary) from baseline to each study visit.</li> </ul> |
| To evaluate disease flare/relapse<br>during and after treatment with<br>mepolizumab SC | <ul> <li>Proportion of subjects who have an IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2-grade improvement during the Treatment and Follow-up Periods.</li> <li>Proportion of subjects who have an increase in EASI score of &gt;=25% from baseline during the Treatment and Follow-up Periods</li> </ul> |
| To characterize the relationship<br>between efficacy and blood eosinophil<br>count | Mean percentage change in EASI score from<br>baseline to each study visit by baseline blood<br>eosinophil count |
| To investigate the pharmacokinetics<br>of mepolizumab in subjects with<br>moderate to severe AD | Plasma concentration of mepolizumab |
| To investigate the pharmacodynamics<br>of mepolizumab in the blood and in<br>AD lesional skin biopsies | <ul> <li>Ratio to baseline in blood eosinophil counts</li> <li>IL-5 levels (serum free and total)</li> <li>Levels of circulating biomarkers in the blood including immunoglobulin (IgE), eosinophilic cationic protein (ECP), and levels of chemokines such as thymus and activation-regulated chemokine (TARC)</li> <li>Gene expression biomarkers in skin biopsies</li> </ul> |
| To describe the effect of mepolizumab<br>SC on Patient reported Outcomes<br>(PROs) | <ul> <li>Change over time in Daily Sign and Symptom<br/>Severity Diary</li> <li>Change over time in Patient Global Impression of<br/>Severity and Patient Global Impression of Change</li> </ul> |

# 2.3. Study Design



| Overview of St | udy Design and Key Features |
|---|---|
| Dosing | • Study Treatment will be administered by SC injection at the Baseline |
| | visit, Week 4, Week 8, and Week 12 (last dose). |
| Time & Events | Refer to Appendix 1: Schedule of Activities |
| Treatment | Subjects will be randomized in 1:1 ratio to receive either Mepolizumab |
| Assignment | 100 mg SC or Placebo SC. |
| Interim | An interim analysis for futility was performed after approximately 50% of |
| Analysis | subjects were randomized and had the opportunity to complete the Week 8 |
| | visit. Futility was evaluated and pre-specified stopping criteria were met |
| | and declared for termination of the study. Further detailed in Section 3.1 |
| Final | Final analysis is planned for subjects who had enrolled into the study prior |
| Analysis | to the termination of the study. |

# 2.4. Statistical Hypotheses / Statistical Analyses

- No formal hypothesis testing is planned.
- The primary objective of this study is to characterize the clinical activity of mepolizumab. A Bayesian approach will be employed to estimate the posterior probability that
  - 1) the IGA response rate for mepolizumab is 40% or greater, and
  - 2) that the improvement over placebo in IGA response rate is at least 15 percentage points.
- Descriptive statistics including point estimates and corresponding 90% confidence interval and 80% credible interval will be provided for efficacy endpoints.

#### 3. PLANNED ANALYSES

# 3.1. Interim Analyses

An interim analysis for futility and to enable future planning was performed after approximately 50% of subjects were randomized and had the opportunity to complete the Week 8 visit. An interim analysis was not conducted to declare early success of the study.

The interim analyses included the following data:

- An assessment of the proportion of subjects who have an IGA score of 0 or 1 and a minimum 2-grade improvement from baseline at Week 8 and later time points
- Assessments of the key secondary endpoint EASI score (change from baseline and percent change from baseline in EASI score)
- Key safety data which included Laboratory and Vital Signs data.

If a subject withdrew at a scheduled visit at which these data were not scheduled to be collected, or if a subject withdrew between scheduled visits, data were slotted to the next visit where the data were scheduled to be collected according to the study flowchart.

The criteria for futility was based on the predictive probability of success at the final analysis, given the data available at the interim analysis.

- If the posterior probability of at least a 15% difference in the IGA response rates between Mepolizumab and Placebo is greater than 70% then the study is declared successful.
- If the predicted probability of success is below the pre-specified threshold of 10%, then the study may stop for futility. i.e.,

**Study Success:** Success=Posterior Probability (difference in Response rates  $\geq 0.15$ )> 70%

**Stop for Futility**: if Probability(Success)< 10%

Steps to calculate the Probability of Success:

- No predictions were made for data at Week 16 based on Week 8 data.
- It was deemed sufficient to use Week 8 as a surrogate for decision making at the interim based on the fact that we would require Mepolizumab to be effective at this earlier timepoint and then maintained out to Week 16.
- Markov-Chain-Monte-Carlo (MCMC) method in SAS was used to derive the posterior distributions response rate between the Mepolizumab treatment group and the placebo group.
  - o From this distribution, a distribution of predicted number of responses post interim was calculated for each treatment group.
  - The observed and predicted number of responders was added together to give a large number of predicted datasets which was analysed using PROC MCMC and the same Bayesian model with non-informative prior as above but with the "observed" final data being a combination of the observed data at the interim and the predicted data from the posterior distribution at the interim.
  - O The posterior probability of the response rate for Mepolizumab meeting the above criteria and the posterior probability of success at the end of the study was calculated and summarised accordingly.
- Convergence diagnostics of MCMC sample was checked using the DIAGNOSTICS option in SAS.

Additional statistical summaries were calculated to enable future planning:

- The 80% credible intervals for the response rate and difference in response rate was presented.
- The predicted posterior probability of at least a 50% response rate on Mepolizumab is greater than 60% was calculated based on observed data at the interim.

Pre-specified stopping criteria for futility were met during this analysis. There were no safety concerns. Study team had therefore terminated this study.

# 3.2. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All participants who had enrolled into the study prior to the termination of the study as defined in the protocol will be part of final analysis.
- 2. All required database cleaning activities have been completed and final database release (DBR) has been declared by Data Management.
- 3. All protocol deviations have been confirmed.
- 4. All criteria for unblinding the randomisation codes have been met.
- 5. Source Data Lock has been declared by Data Management.
- 6. Randomisation codes have been distributed according to RandAll NG procedures.
- 7. Database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Population Definition / Criteria | |
|---|---|---|
| All Screened | All participants who were screened for eligibility | <ul> <li>Study Population</li> </ul> |
| Enrolled | All participants who passed screening and entered the study including randomized participants Note: Screening failures (who never passed screening even if rescreened) and participants screened but never enrolled into the study (Reserve, Not Used) are excluded from the Enrolled population as they did not enter the study. | |
| Intent-to-<br>Treat | <ul> <li>Comprises of all participants who are randomized and who<br/>received at least one dose of study treatment.</li> </ul> | Study Population Ffficacy |
| | <b>Note:</b> This population will be based on the treatment the participants are randomized to. | Efficacy |
| Safety | Comprises of all participants who received at least one dose of a study treatment will be included in the safety population. | Safety |
| | <b>Note:</b> This population will be based on the treatment the participants actually received. | |
| PK | All participants in the Safety population who received the active study treatment and had at least 1 non-missing PK assessment (Non-quantifiable [NQ] values will be considered as non-missing values). | • PK |
| PD | Comprises of all participants in the ITT population who received at least one dose of study treatment and who also have a baseline serum PD measurement and at least one post-treatment serum PD measurement. | • PD |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| Biopsy | Comprises of all participants in the ITT population who have a baseline measurement and who also have at least one post-treatment PD biomarker measurement derived from skin biopsy samples. | Biopsy sub-study |

Refer to Appendix 9: List of Data Displays which details the population used for each display.

Note: If any re-screened participants are randomized and received at least one dose then that subject will be counted in both Screened and ITT Populations.

#### 4.1. Protocol Deviations

Protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be listed.

Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan (10 November 2016 V1 or higher).

- o Data will be reviewed prior to unblinding and freezing the database to ensure all deviations are captured and categorised on the protocol deviations dataset.
- o This dataset will be the basis for the listings of protocol deviations.

A separate listing of all inclusion/exclusion criteria deviations will also be provided. This listing will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

# 5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| RandAll I | RandAll NG Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| 1 | Placebo SC | Placebo SC | 1 |
| 2 | Mepolizumab 100 mg SC | Mepolizumab 100 mg SC | 2 |

#### NOTES:

1. Order represents treatments being presented in TFL

#### 5.2. Baseline Definitions

For all endpoints, the baseline value will be the latest pre-dose assessment. In case of missing pre-dose assessment screening would be considered as baseline. If both are missing, then baseline would be set to missing.

| Parameter | Study Assessments Considered as Baseline | | Baseline Used in<br>Data Display |
|---|---|---|---|
| | Screening [1] | Day 1 (Baseline) | |
| Efficacy Assessments | | | |
| IGA | Χ | X | Day 1 (Baseline) |
| EASI | Х | Х | Day 1 (Baseline) |
| %BSA Affected | Х | Х | Day 1 (Baseline) |
| Daily Sign and Symptom Severity Diary (only for item #1) [2] | Х | X | |
| Patient Global Impression of Severity | | Х | Day 1 (Baseline) |
| Safety Assessments | | | |
| Vital Signs | Х | Х | Day 1 (Baseline) |
| Haematology with differential Clinical Chemistry | Х | Х | Day 1 (Baseline) |
| ECG | Х | | Screening |
| Laboratory Assessments | | · | |
| Immunogenicity (blood samples) | | Х | Day 1 (Baseline) |

<sup>[1]</sup> Screening = 1-2 Wks Prior to Baseline Visit (All Participants).

## 5.2.1. Derivations and Handling of Missing Baseline Data

For untransformed data, change from baseline at each time point is expressed as a difference (value at time point – value at baseline). For log transformed data, change from baseline at each time point is expressed as a ratio (value at time point/value at baseline).

| Definition | Reporting Details |
|---|---|
| Change from Baseline [1] = Post-Baseline Visit Value – Baseline Value | |
| % Change from Baseline [1] = 100 x [(Post-Baseline Visit Value – Baseline) / Baseline] | |
| Ratio to Baseline [2] = Post-Baseline Visit Value/Baseline | |
| [1] If the baseline value is missing the change from baseline derivations will also be missing | |
| [2] Ratio to baseline = Back transformed change from baseline of the loge transformed values | |

# 5.3. Other Considerations for Data Analyses and Data Handling Conventions

Other considerations for data analyses and data handling conventions are outlined in the appendices:

<sup>[2]</sup> Baseline for Daily Sign and Symptom Severity Diary (only for item #1) is based on derivation mentioned in Section 12.2.1

| Section | Component |
|---|---|
| Section 12.2 | Appendix 2: Assessment Windows |
| Section 12.3 | Appendix 3: Study Phases and Treatment Emergent Adverse Events |
| Section 12.4 | Appendix 4: Data Display Standards & Handling Conventions |
| Section 12.5 | Appendix 5: Derived and Transformed Data |
| Section 12.6 | Appendix 6: Reporting Standards for Missing Data |
| Section 12.7 | Appendix 7: Values of Potential Clinical Importance |

# 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Study Population Analyses

The study population analyses will be based on the "Screened", "Enrolled" and "ITT" population, unless otherwise specified.

Study population analyses including analyses of participants' disposition, protocol deviations, demographic and baseline characteristics, prior and concomitant medications, and exposure will be based on GSK Core Data Standards (displays). Details of the planned displays are presented in Appendix 9: List of Data Displays.

## 7. EFFICACY ANALYSES

## 7.1. Primary Efficacy Analyses

#### 7.1.1. Endpoint / Variables

 Proportion of subjects who achieve treatment success defined as an IGA score of 0 or 1 and at least a 2-grade improvement at Week 16

#### 7.1.2. Summary Measure

Posterior mean and median response rate and difference between mepolizumab and placebo and the 80% credible interval for the response rate and the difference in response rate will be presented.

## 7.1.3. Strategy for Intercurrent (Post-Randomization) Events

There are no planned strategies for intercurrent events.

#### 7.1.4. Population of Interest

The primary efficacy analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

#### 7.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays. and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.1.1 will be summarised using descriptive statistics and listed.

#### 7.1.5.1. Statistical Methodology Specification

#### **Endpoint**

 Proportion of subjects who achieve treatment success defined as an IGA score of 0 or 1 and at least a 2-grade improvement at Week 16

#### **Model Specification**

- A non-informative prior will be assumed for the response rate for Mepolizumab and Placebo.
- Markov-Chain-Monte-Carlo (MCMC) method in SAS will be used to derive the posterior distributions for the response rates for Mepolizumab and placebo treatment groups and the difference in response rates between the Mepolizumab and placebo.

#### **Model Checking & Diagnostics**

 Convergence diagnostics of MCMC sample will be checked using the DIAGNOSTICS option in SAS and the alternative method may be used in case convergence is not achieved.

#### **Model Results Presentation**

- Posterior mean and median response rate and difference between mepolizumab and placebo and the 80% credible interval for the response rate and the difference in response rate will be presented.
- The posterior probability that the IGA response rate for mepolizumab is 40% or greater and that the improvement over placebo is at least 15 percentage points will be calculated.

#### **Sensitivity and Supportive Analyses**

There are planned sensitivity or supportive analyses.

# 7.2. Secondary Efficacy Analyses

# 7.2.1. Endpoint / Variables

- EASI Score
- IGA Response rate

# 7.2.2. Summary Measure

- Mean Change from baseline & percentage change from baseline EASI score to each visit
- Proportion of subjects with an IGA score of 0 or 1 and at least a 2-grade improvement from baseline to each visit

## 7.2.3. Strategy for Intercurrent (Post-Randomization) Events

There are no planned strategies for intercurrent events.

## 7.2.4. Population of Interest

The secondary efficacy analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

# 7.2.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 7.2.1 will be summarised using descriptive statistics and listed.

#### 7.2.5.1. Statistical Methodology Specification

There will be no planned statistical analysis.

# 7.3. Exploratory Efficacy Analyses

## 7.3.1. Endpoint / Variables

- At least 50% and 75% improvement in EASI score from baseline
- Total body surface area (% BSA)
- Weekly average of daily itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary)
- IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2-grade improvement during the Treatment and Follow-up Periods.
- Increase in EASI score of >=25% from baseline during the Treatment and Follow-up Periods.
- EASI score by baseline blood eosinophil count
- Daily Sign and Symptom Severity Diary
- Patient Global Impression of Change
- Patient Global Impression of Severity
- Clinician Global Impression of Change

#### 7.3.2. Summary Measure

- Proportion of subjects with ≥50% improvement (i.e., -50% percent change from baseline) in EASI from baseline to each visit.
- Proportion of subjects with ≥75% improvement (i.e., -75% percent change from baseline) in EASI from baseline to each visit.
- Mean change in weekly average of daily itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary) from baseline to each visit.

- Mean Percentage Change in EASI score from Baseline to each visit by baseline blood eosinophil count quartiles.
- Only listings will be presented for [1] IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2-grade improvement during the Treatment and Follow-up Periods, [2] Increase in EASI score of >=25% from baseline during the Treatment and Follow-up Periods. [3] Total body surface area (% BSA), [4] Daily Sign and Symptom Severity Diary, [5] Patient Global Impression of Change and Severity and [6] Clinician Global Impression of Change endpoints.

## 7.3.3. Strategy for Intercurrent (Post-Randomization) Events

There are no planned strategies for intercurrent events.

#### 7.3.4. Population of Interest

The exploratory efficacy analyses will be based on the "Intent-To-Treat" population, unless otherwise specified.

#### 7.3.4.1. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

Unless otherwise specified, endpoints defined in Section 7.3.1 will be summarised using descriptive statistics and listed.

#### 7.3.4.2. Statistical Methodology Specification

There will be no statistical analysis, only descriptive statistics will be presented.

#### 8. SAFETY ANALYSES

The safety analyses will be based on the "Safety" population, unless otherwise specified.

# 8.1. Adverse Events Analyses

Adverse events analyses including the analysis of adverse events (AEs), Serious (SAEs) and other significant AEs will be based on GSK Core Data Standards. The details of the planned displays are provided in Appendix 9: List of Data Displays.

## 8.2. Adverse Events of Special Interest Analyses

Adverse events of special interest (AESIs) are adverse events associated with the identified and potential risks of mepolizumab. AESIs reported by the investigator as anaphylaxis reactions, systemic reactions (further categorised by the investigator as either allergic (type I hypersensitivity) or other systemic reactions) and local injection site reactions are collected via targeted eCRF within the study.

The AESIs of opportunistic infections, malignancies, serious CVT events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset; created based on the latest version of the MedDRA dictionary available at the time of database freeze for this study.

Separate summary tables showing the number and percent of subjects with type of AESI, broken down by preferred term will be created if at least one event is reported for an AESI category. For each type of AESI a profile summary table will be produced containing information including, but not limited to, the number of occurrences of the event, event characteristics, time to onset, intensity, outcome and action taken if more than one event is reported for an AESI category.

Listings of AESIs identified by the investigator as anaphylaxis, allergic (type I hypersensitivity), other systemic reactions and local injection site reactions, opportunistic infections, malignancies, serious CVT events and serious ischemic events if more than one event is reported under each AESI category.

The details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK data standards and statistical principles.

# 8.3. Clinical Laboratory Analyses

Laboratory evaluations including the analyses of Chemistry laboratory tests, Haematology laboratory tests and liver function tests will be based on GSK Core Data Standards. A scatter plot of maximum ALT vs baseline ALT, and maximum ALT vs total bilirubin will be produced. In addition, if any liver stopping or liver monitoring events occur during the study, then only listing of liver monitoring/stopping event reporting and hepatobiliary laboratory abnormalities will be produced. The details of the planned displays are in Appendix 9: List of Data Displays.

# 8.4. Other Safety Analyses

The analyses of non-laboratory safety test results including ECGs and vital signs will be based on CDISC Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays.

#### 8.4.1. ECG

All sites used a standardised ECG equipment provided by a centralised external vendor. A central ECG reader was used. The site and vendor provided ECG interpretation, while the site differentiates between "Abnormal – Not Clinically Significant and Abnormal – Clinically significant", the vendor only specifies 'Abnormal'. There are differences between the site vs vendor interpretations (i.e. the site interpretation = abnormal vs vendor = normal and site = normal vs vendor = abnormal).

As site interpretations also take into consideration assessment from investigators of patients, the site interpretations will be used for summaries (i.e. even though for patients, vendor = abnormal vs site = normal) but both the site and vendor interpretations will be listed.

Actual and change from baseline QTcF category values will be summarized for each visit. Actual QTcF value is categorized as: <=450, >450 to <=480, >480 to <=500, and >500. Change from baseline QTcF value is categorized as: <=30, >30 to  $\le60$  and >60. In addition, listing will be produced for subject meeting the criteria of actual QTcF >500 msec or change from baseline >60 msec.

# 8.5. Immunogenicity Analyses

Immunogenicity analyses will be based on GSK Core Data Standards, unless otherwise specified. The details of the planned displays are presented in Appendix 9: List of Data Displays in Section 12.9.6.

An immune response to a therapeutic drug can lead to generation of anti-drug antibodies within the blood. For the immunogenicity assessment, two types of antibody assays will be performed, a binding antibody assay and a neutralizing antibody assay.

For the binding antibody assay, there will be three testing steps: screening, confirmation and titration. The screening assay produces a result of positive or negative relative to a screening cut point. Positive samples continue with the confirmation assay, which also produces a result of positive or negative relative to a confirmation cut point. For samples with a positive confirmation result, a titre value will also be obtained to quantify the degree of binding in a titration assay and the sample will be characterized as positive for the binding antibodies. Subjects who test positive for the binding antibody assay, will be tested in the neutralizing antibody assay, which also reports results as positive or negative.

Subjects will be categorized as negative or positive and positive binding antibody will be further categorized as transient positive or persistent positive at each visit and for anytime post baseline visit. Summary statistics for titer results will also be included for anytime post baseline visit.

A summary of adverse events by highest post-baseline binding antibody result will be produced. A summary of treatment emergent positive confirmation binding ADA assay results in the subset of subjects who did not have a positive confirmation binding ADA assay result prior to the dosing of study treatment will also be presented.

Neutralizing antibody assay results will be summarised by visit and will also be summarised by category (positive or negative). For anytime post baseline visit, highest result will be used, i.e. according to the following hierarchy: ADA result will be Persistent Positive > Transient Positive > Negative, NAB result will be Positive > Negative and highest titer value. A listing of all immunogenicity data will also be provided.

#### 9. PHARMACOKINETIC ANALYSES

## 9.1. Exploratory Pharmacokinetic Analyses

## 9.1.1. Endpoint / Variables

Plasma concentration of mepolizumab.

### 9.1.1.1. Drug Concentration Measures

Mepolizumab plasma concentrations will be summarised and listed by nominal time. Standard summary statistics will be calculated.

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 12.5.3 Reporting Standards for Pharmacokinetic).

#### 9.1.1.2. Derived Pharmacokinetic Parameters

As a result of study termination, there will be no derivation of Pharmacokinetic Parameters for this study.

#### 9.1.2. Summary Measure

There is no treatment comparison in this study since only one active study treatment was administered. Mepolizumab plasma Concentrations will be summarised descriptively.

#### 9.1.3. Population of Interest

The exploratory pharmacokinetic analyses will be based on the "Pharmacokinetic" population, unless otherwise specified.

#### 9.1.4. Strategy for Intercurrent (Post-Randomization) Events

Missing concentrations and concentrations below the limit of quantification of the assay will be handled as described in Guidance Document GUI 51487.

#### 9.1.5. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Core Data Standards and statistical principles.

Unless otherwise specified, endpoints / variables defined in Section 9.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

#### 10. PHARMACODYNAMIC AND BIOMARKER ANALYSES

# 10.1. Exploratory Pharmacodynamic and Biomarker Analyses

#### 10.1.1. Endpoint / Variables

| Endpoint | Parameters |
|---|---|
| Biomarker(s) / | Blood Sample: Eosinophil counts |
| Pharmacodynamic Markers | Blood Sample: IL5 levels (serum free and total) |
| Novel Biomarkers – Skin Biops | sy Sub-study & Serum Biomarkers |
| RNA Transcriptome Research | • N/A |
| (Cancelled) | |
| RNA Expression Research of a | Gene expression biomarkers in skin biopsies |
| Subset of RNA Species [1] | |
| Protein Levels of Biomarkers in | Total IgE, eosinophil cationic protein (ECP) and |
| Serum [2] | chemokines Eotaxin-1, Eotaxin-3, TARC, MCP4 |
| [1] Epistem will be providing a report to be include in the CSR. | |
| [2] MDC was dropped as an analyte due to assay issues) | |

## 10.1.2. Summary Measure

- Geometric Means for ratio to baseline in blood eosinophil counts and for absolute blood eosinophil count at each visit.
- Only listings will be presented for biomarker endpoints.

#### 10.1.3. Population of Interest

The pharmacodynamics and biomarker analyses will be based on the "Safety", "Pharmacodynamic" and "Biopsy" populations, unless otherwise specified.

Safety population will be used for summarizing blood eosinophil counts. Biopsy population will be used for skin biopsy. Pharmacodynamic population will be used for remaining endpoints.

#### 10.1.4. Statistical Analyses / Methods

Details of the planned displays are provided in Appendix 9: List of Data Displays and will be based on GSK Data Standards and statistical principles.

Unless otherwise specified, endpoints/variables defined in Section 10.1.1 will be summarised using descriptive statistics, graphically presented (where appropriate) and listed.

# 10.1.4.1. Statistical Methodology Specification

#### **Endpoint**

Ratio to baseline blood eosinophil counts (Note: from standard haematology assessments)

### **Model Specification**

- Mixed Models Repeated Measures (MMRM) analysis.
- The analysis will include all measurements at scheduled visits
- Terms in the model:
- Response: Ratio to Baseline Blood eosinophil count (loge transformed prior to analysis) (see Appendix 5: Derived and Transformed Data, Section 12.5.6).
  - Categorical: Treatment group, Visit.
  - Continuous/covariate: Baseline blood eosinophil count.
  - Interaction: Treatment group\*Visit.
  - Repeated: Visit.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used. An unstructured covariance structure for the R matrix will be used by specifying 'type=UN' on the REPEATED line.

# **Model Checking**

 Distributional assumptions underlying the model used for analysis will be examined by obtaining a normal probability plot of the residuals and a plot of the residuals versus the fitted values (i.e. checking the normality assumption and constant variance assumption of the model respectively) to gain confidence that the model assumptions are reasonable.

#### **Model Results Presentation**

 The results of the analysis from the MMRM model will be presented for each visit as LS Geometric Mean (SE), LS Geometric Mean Ratio to Baseline (95% Confidence Interval) for each treatment group, Geometric Treatment Ratio (Mepolizumab/Placebo) and corresponding 95% Confidence Interval.

#### **Sensitivity and Supportive Analyses**

There are no planned sensitivity or supportive analyses.

# 11. REFERENCES

GlaxoSmithKline Document Number 2015N268158\_02, Study ID 205050, A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Investigate the Efficacy and Safety of Mepolizumab Administered Subcutaneously in Subjects with Moderate to Severe Atopic Dermatitis. Effective Date: 22-JUN-2017.

# 12. APPENDICES

# 12.1. Appendix 1: Schedule of Activities

Time and Events Table: Pre-Screening and Screening

| Period: | Pre-Screening ar | nd Screening | Period |
|---|---|---|---|
| | | | Notes |
| Visits: | Pre-Screening | Screening | |
| | Up to 4 wks<br>prior to<br>Screening Visit | 1 to 2 wks<br>prior to<br>Day 1<br>Baseline<br>Visit | Individual Pre-Screening and Screening Visits will be conducted for subjects who have used prohibited medications or non-drug therapies and need to fulfil the prohibited medications period prior to the Screening Visit (See Table 1). For these subjects, the Pre Screening Visit will be completed up to 4 weeks prior to the Screening Visit. After requirements regarding previous use of prohibited medication and non-drug therapies are met (See Table 1), the Screening Visit will be completed. The Screening visit will be completed up to 2 weeks prior to the Baseline visit. Assessments for Pre-screening and Screening Periods will be combined into one Screening Visit for subjects who meet prohibited medications or non-drug therapies criteria in Table 1 at entry (total time to complete the combined assessments= 1 to 2 weeks prior to Baseline). The period between the Screening Visit and Baseline Visit may be extended beyond 2 weeks, if needed, to obtain the results of all screening laboratory assessments. |
| Procedure | | | |
| Informed consent | PS | Si X | Obtain informed consent prior to study participation. See Section 4.2.1 and Table 1 notes. |
| Demography | PS | | |
| Fitzpatrick Skin Type Classification | PS | g y | |
| Inclusion/exclusion criteria | PS | S | and the same of th |
| Medical history/Medical conditions | PS | s | Includes drug and alcohol usage, smoking history, cardiovascular medical history, and<br>family history of premature cardiovascular disease. |
| Safety Assessments | | | |
| Vital Signs | | S | See Section 7.4.4. |
| Concomitant medications | PS | S | The subject must apply the same non-prescription, non-medicated emollient twice daily for<br>the 7 consecutive days immediately prior to the Baseline visit. On study visit days,. |
| | | | emollient must not be applied within the 2-hour period preceding the study visit. If<br>emollient is applied <2 hours prior to the visit, wait ≥2 hours after application to perform<br>study procedures. See Section 6.10.1 |
| Serious Adverse Events (SAEs) | PS | S | Record SAEs related to study participation or to a GSK product from the time a subject<br>consents to participate in the study up to and including any follow-up contact. AEs will be<br>collected from the start of study treatment until the follow-up contact (Section 7.4.1.1). |
| ECG | | S | |
| Laboratory Assessments | Note: Results of | all laboratory | assessments must be available prior to randomization |
| HBsAG and hepatitis C antibody | PS | | Not required if test otherwise performed within 3 months prior to first dose of study treatment. |
| Pregnancy test (urine) | PS | S | Females of reproductive potential. If urine pregnancy test is positive, collect serum hCG (central laboratory). See Section 7.4.2 and Appendix 7 for reporting requirements. |
| FSH and estradiol | PS | | Females, if needed to confirm postmenopausal status (See Section 5.1). |
| Hematology with differential | | S | |
| Clinical Chemistry | | S | |
| Parasitic screening | | S | Parasitic screening is only required in countries with high-risk or for subjects who have<br>visited high-risk countries in the past 6 months. Sites should use local laboratories.<br>Selection of tests will be at the investigator's judgment. |
| Efficacy Assessments and Patient-Re | eported Outcomes | | Variation of the control of the cont |
| Investigator's Global Assessment | | S | See Section 7.3 and SRM for rater requirements. Regional assessment. Total % BSA affected will be auto-calculated within the eCRF. The |
| % BSA affected | | 8 | total %BSA score from the eCRF will be utilized to confirm inclusion criteria. See Section 7.3 and SRM for rater requirements. |
| EASI | | 8 | % BSA affected will be utilized to calculate the EASI score. The EASI score will be auto-<br>calculated within the eCRF. The EASI score from the eCRF will be utilized to confirm<br>inclusion criteria. See Section 7.3 and SRM for rater requirements |
| Daily Sign and Symptom Severity<br>Diary (electronic) | | S | To be completed by the subject every evening before 12:00 AM (midnight). If subject fails screening and does not continue in the study, the subject will return the electronic device to the site. (See SRM for quidance). |

# Time and Events Table: Baseline through Follow-up Period

| Period: | Treatment | | | | | Follow-up<br>Period | | Notes |
|---|---|---|---|---|---|---|---|---|
| | N 32 20 2 | | | Post-Tx<br>Visit 1<br>4 wks after<br>last dose | Post-Tx<br>Visit 2<br>8 wks after<br>last dose | Early | Perform procedures in the order listed in Section 7. Early WD visit: same procedures apply both to subjects discontinuing treatment but continuing with Post-Tx visits and to subjects withdrawing from the study. | |
| Day/Week: | Day 1<br>Baseline | Wk 4 | Wk 8 | Wk 12 | Wk 16<br>(No IP<br>dose) | Wk 20<br>(No IP<br>dose) | WD | |
| Window (days): | | ±3 | ±3 | ±3 | ±3 | ±3 | | |
| Procedure | | | 0 0 | | | | | |
| Inclusion/exclusion criteria | BL | | | | | | | |
| Randomization (IVRS) | BL | | | | | i i | | |
| Safety Assessments | N: 17 | | | 4 4 | | : 7 | • | ů. |
| Physical examination, height, weight | BL | | | | - 6 | 20 | EW | Perform/obtain pre-dose on dosing days. See Section 7.4.3. |
| Vital signs | BL | 4 | 8 | 12 | 16 | 20 | EW | Obtain pre-dose on dosing days. See Section 7.4.4. |
| ECG | | 4 | | | 16 | | EW | Obtain pre-dose at Week 4. Unscheduled ECGs may also be performed as clinically indicated during the study. |
| Concomitant medications | BL | 4 | 8 | 12 | 16 | 20 | EW | preceding the study visit. If emollient is applied <2 hours<br>prior to the visit, wait ≥2 hours after application to perform<br>study procedures. |
| Adverse events | BL | 4 | 8 | 12 | 16 | 20 | EW | Collect AEs from the start of study treatment until the follow<br>up contact. Record SAEs related to study participation or to<br>a GSK product from the time a subject consents to<br>participate in the study up to and including any follow-up<br>contact (Section 7.4.1.1). |
| Laboratory Assessments | Note: | Labs a | re col | lected p | re-dose on | dosing days | (inclu | des blood draws, skin biopsies, and pregnancy testing) |
| Genetic sample- pre-dose | BL | | | | | | | Subject participation is voluntary. Additional informed consent is required. |
| Hematology with differential | BL | 4 | 8 | 12 | 16 | 20 | EW | Total WBC, absolute eosinophil count, and differential (%) will be blinded from the Baseline visit until the end of the study. |
| Clinical Chemistry | BL | 4 | 8 | 12 | 16 | | EW | |
| Pregnancy test (urine) | BL | 4 | 8 | 12 | 16 | 20 | EW | Females of reproductive potential. If urine pregnancy test is<br>positive, collect serum hCG (central laboratory). See Section<br>7.4.2 and Appendix 7 for reporting requirements. |
| Pharmacokinetic blood sample | | 4 | 8 | 12 | 16 | 20 | EW | Results will be blinded during the study. |
| Blood sample for immunogenicity | BL | 4 | | | 16 | 20 | | Results will be blinded during the study. |
| Serum IL-5 | BL | 4 | | | 16 | 20 | EW | Results will be blinded during the study. |
| Serum sample for biomarkers | BL | 4 | 8 | 12 | 16 | | 10000 | Results will be blinded during the study. |
| Skin biopsy sub-study-<br>pre-identified study centers only | BL | 4 | | | | | | Subject participation is voluntary. Additional informed consent is required. Results will be blinded during the study Collect 1 lesional sample (from chronic lesion) and 1 non-lesional sample at each visit. |
| Efficacy Assessments and Patient-Re | ported Ou | tcome | s | | | | | Assessment of the second secon |
| Patient Global Impression of Change | | 4 | 8 | 12 | 16 | | EW | Complete pre-dose prior to other assessments or evaluation by the investigator. |

| Efficacy Assessments and Patient-Re | ported Ou | itcome | 8 | - 1 | | | | IA |
|---|---|---|---|---|---|---|---|---|
| Patient Global Impression of Severity | BL | 4 | 8 | 12 | 16 | 20 | EW | Complete pre-dose prior to other assessments or evaluation<br>by the investigator. |
| Daily Sign and Symptom Severity<br>Diary (electronic) | <del>(</del> | | EW | To be completed by the subject every evening before<br>12:00 A.M.(midnight) during the Treatment and Follow-up<br>Periods. Site personnel will review subject compliance with<br>the diary at each visit. | | | | |
| Investigator's Global Assessment | BL | 4 | 8 | 12 | 16 | 20 | EW | Complete pre-dose. See Section 7.3 and SRM for rater requirements. |
| % BSA affected | BL | 4 | 8 | 12 | 16 | 20 | EW | Complete pre-dose. Regional assessment. Total % BSA affected will be auto-calculated within the eCRF. See Section 7.3 and SRM for rater requirements |
| EASI | BL | 4 | 8 | 12 | 16 | 20 | EW | Complete pre-dose. % BSA affected from each visit will be utilized to calculate the EASI score at each visit. The EASI score will be auto-calculated within the eCRF. See Section 7.3 and SRM for rater requirements |
| Clinician Global Impression of Change | | 4 | 8 | 12 | 16 | | EW | Complete pre-dose. See Section 7.3. and SRM for rater requirements |
| Investigational Product and Other Stu | dy Treatn | nent | 01 1 | | 12. 33 | 1 10 | | |
| Mepolizumab or Placebo<br>Administration | BL | 4 | 8 | 12 | No IP dose | No IP dose | | See Section 6.1 and Section 6.1.1 for study treatment administration details. Observation of subject required for 1 hour after administration of study treatment. See Section 6.1.2. Postponement of study treatment and visit assessment is required during course of antibiotic, antiviral or antifungal treatment for acute infection. Postponed doses can be administered no further than 2 weeks after the original scheduled dose (See Section 5.4.3). |

#### Time and Events Table: Unscheduled Visit for Flare/Relapse

| Period: | Treatment<br>and Follow-<br>up | |
|---|---|---|
| 3 | 9 9 | Notes |
| Week: | Unscheduled | <ul> <li>This visit is for subjects who experience AD flare/relapse between scheduled study visits. See Section 4.2.4.</li> <li>In the case of flare/relapse with intolerable AD symptoms where the use of prohibited medication is required (See Table 1), the subject will be permanently withdrawn from treatment.</li> </ul> |
| | | If the subject permanently discontinues study treatment or withdraws from the study, the procedures and visits described in Section 5.4 and Table 3 will apply. Perform procedures in the order listed in Section 7. |
| Window (days): | +5 | Visit window is from the time the subject notifies the site staff of potential AD flare/relapse. |
| Procedure | ** | |
| Safety Assessments | | 2 |
| Physical examination,<br>height, weight | U | To be performed only if needed, based on the investigator's judgment. |
| Vital signs | U | See Section 7.4.4: |
| Concomitant medications | U | ac comment was |
| Adverse events U | | See Appendix 11. The disease under study (AD) or expected<br>progression, signs, or symptoms of AD do not meet the<br>definition of AE unless the worsening is more severe than<br>expected for the subject's condition. |
| Laboratory Assessments | | |
| Hematology with U | | Total WBC, absolute eosinophil count, and differential (%) will<br>remain blinded. |
| Clinical Chemistry | U | Performed only if needed, based on investigator's judgment. |
| Efficacy Assessments and | Patient-Report | |
| Daily Sign and Symptom<br>Severity Diary (electronic) | U | To be completed the by subject in the evening. |
| Investigator's Global<br>Assessment | U | 1/2 |
| % BSA affected | U | Regional assessment. Total % BSA affected will be auto-<br>calculated within the eCRF. See Section 7.3 and SRM for rat<br>requirements. |
| EASI U | | % BSA affected from each visit will be utilized to calculate the<br>EASI score at each visit. The EASI score will be auto-<br>calculated within the eCRF. See Section 7.3 and SRM for rater<br>requirements. |

Abbreviations: AEs= adverse events; BSA= body surface area; EASI= Eczema Area and Severity Index; FSH= follicle stimulating hormone; HBsAG= hepatitis B surface antigen; SAEs= serious adverse events; SRM=Study Reference Manual. AD= atopic dermatitis; EASI= Eczema Area and Severity Index; WBC= white blood cell; WD=withdrawal; IL-5= interleukin-5; Tx= Treatment; Wk=Week; wks=weeks

# 12.2. Appendix 2: Assessment Windows

Clinic visits are scheduled to take place as specified in the protocol. Unscheduled visit will be excluded from analyses on any population. For all clinic visits, nominal visit days and times will be used for reporting; for example, if a subject recorded value on the Week 4 visit that were made on Week 3 of treatment, they will be presented as Week 4 values.

If a subject withdraws at a scheduled visit, and these data were scheduled to be collected at that visit, the data will be summarised and analysed (as appropriate) together with data from subjects who did not withdraw. If a subject withdraws at a scheduled visit at which these data were not scheduled to be collected, or if a subject withdraws between scheduled visits, data will be slotted to the next visit where the data was scheduled to be collected according to the study flowchart. The protocol visits windows of  $\pm 3$  days should be applied to the assignment of withdrawal visits, so that if a subject withdraws within the appropriate number of days from the last visit where that data was scheduled to be collected, they would get that data slotted to that visit and otherwise the data will be slotted to the next scheduled visit.

The early withdrawal visit will then be re-labelled as the corresponding visit. The same approach will be followed to Post Treatment 1 and Post Treatment 2 visits.

If there is more than one assessment associated with a particular visit interval, then the latest assessment will be used for summary tables and analyses. Where two or more findings (e.g. ECG (i.e. site interpretations will be used), laboratory data) slot to the same visit interval, the most 'abnormal' results will be used, i.e. according to the following hierarchy: Abnormal-Clinically Significant > Abnormal – not clinically significant > Normal.

## 12.2.1. Definitions of Assessment Windows for Analyses

The daily itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary) is recorded daily and will be averaged for every week.

The 7-days average score will be calculated as:

# $\Sigma$ (Daily itch/pruritus NRS score in 7 days)

Total numer of days Daily itch/pruritus NRS score is recorded in 7 days \*

- If a subject is missing more than 3 daily itch/pruritus NRS scores out of the 7 days, then the average NRS score for that week will be recorded as missing.
- 7-days average score for baseline visit will be calculated based on 7 days prior to the day of dosing (i.e., from Day -7 to Day -1).
- 7-days average score for Week 1 visit will be 7 days after the day of dosing (i.e., from Day 1 to Day 7).
- Similarly, for Week 2 (from Day 8 to Day 14) and henceforth till Week 20.

# 12.3. Appendix 3: Study Phases and Treatment Emergent Adverse Events

## 12.3.1. Study Phases

Safety assessments and events will be classified according to the time of occurrence relative to the first dose of investigational product.

The on-treatment phase for the presentation of exposure, adverse event and concomitant medications is defined as being from the day of the first administration to the day of the last administration of study treatment + another 28 days inclusive.

| Treatment Phase | Definition |
|---|---|
| Pre-Treatment | Date < IP start date |
| On-Treatment | Event onset date is on/after IP start date & on/before IP stop date + 28 days |
| | (IP Start Date ≤ Date ≤ IP Stop Date + 28 days) |
| Post-Treatment | Event onset date is after the IP stop date + 28 |
| | (Date > IP stop date + 28) |
| IP = Investigational | Product = Study Treatment |

#### 12.3.1.1. Study Phases for Efficacy Assessments

Efficacy assessments and events will be classified according to the time of occurrence relative to the study periods defined below:

| Period | Definition |
|---|---|
| Study Treatment Period | Date ≤ Week 16 date (or date of withdrawal from the study, if prior to Week 16) |
| Follow-up Period | Week 16 date < Date ≤ Week 20 date (or date of withdrawal from the study, if |
| | between Week 16 and 20) |

#### 12.3.2. Treatment Emergent Flag for Adverse Events

| Flag | Definition |
|---|---|
| Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date. (plus |
| Emergent | 28 days) |
| | (Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 28) |

#### NOTES:

- If the study treatment stop date is missing, then the AE will be considered to be On-Treatment.
- Time of study treatment dosing and start/stop time of AEs should be considered, if collected.

# 12.4. Appendix 4: Data Display Standards & Handling Conventions

# 12.4.1. Reporting Process

| Software | |
|---|---|
| The currently supported versions of SAS software 9.4 or higher will be used. | |
| Reporting Area | |
| HARP Server | : uk1salx00175.corpnet2.com |
| HARP Compound | : sb240563\mid205050\final_02 |
| QC Spreadsheet | : sb240563\mid205050\ final_02\documents |
| Analysis Datasets | |

- Analysis datasets will be created according to CDISC standards (SDTM IG Version 3.1.3 & ADaM IG Version 1.0].
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for SAC.

#### 12.4.2. Reporting Standards

#### General

 The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated (IDSL Standards Location:

https://spope.gsk.com/sites/IDSLLibrary/SitePages/Home.aspx):

- 4.03 to 4.23: General Principles
- 5.01 to 5.08: Principles Related to Data Listings
- 6.01 to 6.11: Principles Related to Summary Tables
- 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected, unless otherwise stated.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days
    on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.

| Unscheduled Visits | |
|---|---|
| Unscheduled visit | Unscheduled visits will not be included in summary tables and/or figures. |
| All unscheduled v | All unscheduled visits will be included in listings. |
| Descriptive Summar | y Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| <b>Graphical Displays</b> | |
| Refer to IDSL Sta | tistical Principals 7.01 to 7.13. |

# 12.4.3. Reporting Standards for Pharmacokinetic

| Pharmacokinetic Concentration Data | |
|---|---|
| Descriptive Summary | Refer to IDSL PK Display Standards. |
| Statistics, Graphical | Refer to IDSL Statistical Principle 6.06.1. |
| Displays and Listings | Note: BLQ Concentration values will be imputed as per GUI_51487 for descriptive |
| | summary statistics and summarized graphical displays only. |

# 12.5. Appendix 5: Derived and Transformed Data

#### 12.5.1. General

#### **Multiple Measurements at One Analysis Time Point**

- If there are two values within a time window (as per Section 12.2.1) then the latest assessment will be used.
- Participants having both High and Low values for Normal Ranges at any post-baseline visit for safety parameters will be counted in both the High and Low categories of "Any visit post-baseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### **Study Day**

- Calculated as the number of days from Randomization Date:
  - Ref Date = Missing
- → Study Day = Missing
- Ref Date < Randomization Date → Study Day = Ref Date Randomization Date</li>
- Ref Data ≥ Randomization Date → Study Day = (Ref Date Randomization Date) + 1

# 12.5.2. Study Population

#### **Extent of Exposure**

- Number of days of exposure to study drug will be calculated based on the formula: Duration of Exposure in Days = (Treatment Stop Date – Treatment Start Date) + 29
- Participants who were randomized but did not report a treatment start date will be categorised as having zero days of exposure.
- On-treatment phase will be calculated based on the formula: On-Treatment Phase = (Treatment Stop Date – Treatment Start Date) + 29

## 12.5.3. **Efficacy**

#### **Efficacy**

#### **Investigators Global Assessment (IGA)**

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

- A Responder is defined as a subject who has an IGA score of 0 or 1 and a minimum 2-grade improvement from baseline. This is calculated for each study visit.
- As per protocol, a non-responder imputation will be used for all early withdrawal subjects where

#### **Efficacy**

- subject's data will be imputed as a Non-Responder for all post withdrawal visits. This imputation will be used for summary and analysis table for primary and secondary endpoints.
- The observed IGA score classifications will be used for each visit. For all early withdrawal subjects the data from Post-Treatment 1/Post-Treatment 2/Early Withdrawal visits will be slotted using the algorithm detailed in Section 12.2
- AD flare/relapse for IGA is defined as IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2- grade improvement from the baseline.

### **Body Surface Area**

| Body Region | % Involvement (0-100% each area) | % Involvement x Proportionality Multiplier | Regional % BSA<br>Involvement |
|---|---|---|---|
| Head and neck | | x 0.1 | |
| Upper extremities | | x 0.2 | |
| Trunk | | x 0.3 | |
| Lower extremities | | x 0.4 | |

#### **EASI**

CCI - This section contained Clinical Outcome Assessment data collection questionnaires or indices, which are protected by third party copyright laws and therefore have been excluded.

- The observed EASI data will be used for each visit. For all early withdrawal subjects, data from Post-Treatment 1/Post-Treatment 2/ Early Withdrawal visits will be slotted using the algorithm detailed in Section 12.2.
- AD flare/relapse for EASI is defined as increase in EASI score of ≥25% from Baseline.
### 12.5.4. Safety

#### **Adverse Events of Special Interest**

- Section 8.2: Adverse Events of Special Interest Analyses provides a full list of AEs of special interest for this compound. AESIs of anaphylaxis reactions, systemic reactions, and local injection site reactions are collected via targeted eCRF.
- The AESIs of opportunistic infections, malignancies, serious CVT events and serious ischemic events will be identified from a list of relevant preferred terms maintained within a project level reference dataset; created based on the latest version of the MedDRA dictionary available at the time of database freeze for this study (See Program Safety Analysis Plan for additional details).

### **Laboratory Parameters**

- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Decimal Points = '< x' becomes x 0.01</p>
  - Example 2: 1 Decimal Point = '> x' becomes x + 0.1
  - Example 3: 0 Decimal Points = '< x' becomes x 1

### Immunogenicity (Binding Antibody Assay Results)

- Positive binding antibody assay results are to be categorised as transient positive or persistent positive accordingly to the following definitions:
- For all post-baseline visits, other than final study assessment
  - Transient positive = a single positive immunogenic response at a visit, where the previous visit was negative
  - Persistent positive = a positive immunogenic response at a visit, where the previous visit was also positive
- For the final assessment:
  - Any positive response will be considered a persistent response, regardless of the status at the previous visit

#### 12.5.5. Pharmacokinetic

There will be no derivation of Pharmacokinetic Parameters for this study.

### 12.5.6. Pharmacodynamic and Biomarker

### **Pharmacodynamic**

### **Blood Eosinophils**

- Blood eosinophil counts will be log transformed (loge) prior to analysis.
- For the log transformation values of 0 GI/L will be imputed to a value of minimum for all non-missing results/2.

## 12.6. Appendix 6: Reporting Standards for Missing Data

### 12.6.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as if he/she receives all planned doses of study treatment and completes the Week 16 (Post-Treatment 1) and Week 20 (Post-Treatment 2) visits.</li> <li>Withdrawn subjects were not replaced in the study.</li> </ul> |
| | <ul> <li>All available data from participants who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> <li>Withdrawal visits will be slotted as per Appendix 2: Assessment Windows</li> </ul> |

## 12.6.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated using a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any participants excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 12.6.2.1. Handling of Missing and Partial Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 3: Study Phases and Treatment Emergent Adverse Events.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop</li> </ul> </li> </ul> |
| | date of study treatment; in this case the study treatment stop date will be used. |
| | Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

# 12.7. Appendix 7: Values of Potential Clinical Importance

## 12.7.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Age | Clinical Concern Range | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| Hematocrit | Ratio of 1 | 12+ | 0.201 | 0.599 |
| Hemoglobin | G/L | 12+ | 71 | 199 |
| Platelet Count | GI/L | 1+ | 31 | 1499 |
| While Blood Cell Count (WBC) | GI/L | 12+ | 1.1 | |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Age | Clinical Concern Range | |
| | | Category | Low Flag (< x) | High Flag (>x) |
| ALT | U/L | 3-12 | | >143 (and Total<br>Bilirubin >43) |
| | U/L | 13+ | | >239 (and Total<br>Bilirubin >43) |
| Calcium | mmol/L | 3+ | 1.50 | 3.24 |
| Glucose | mmol/L | 1+ | 2.2 | 27.8 |
| Potassium | mmol/L | 3+ | 2.8 | 6.5 |
| Sodium | mmol/L | 0+ | 120 | 160 |

| Possible Hy's Law Cases | | | |
|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range |
| ALT, Bilirubin | | | ALT ≥ 3xULN and Bilirubin ≥ 2xULN (>35% direct) |
| ALT, INR | | | ALT ≥ 3xULN and INR > 1.5 |

## 12.7.2. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | Absolute | | |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 12.8. Appendix 8: Abbreviations & Trade Marks

## 12.8.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AESI | Adverse Events of Special Interest |
| AIC | Akaike's Information Criteria |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| DBF | Database Freeze |
| DBR | Database Release |
| DOB | Date of Birth |
| DP | Decimal Places |
| EASI | Eczema Area and Severity Index |
| eCRF | Electronic Case Record Form |
| ECP | Eosinophilic Cationic Protein |
| EASI | Eczema Area and Severity Index |
| EMA | European Medicines Agency |
| FDA | Food and Drug Administration |
| FDAAA | Food and Drug Administration Clinical Results Disclosure Requirements |
| GSK | GlaxoSmithKline |
| IA | Interim Analysis |
| ICH | International Conference on Harmonization |
| IDSL | Integrated Data Standards Library |
| IGA | Investigator's Global Assessment |
| IGE | Immunoglobulin |
| ITT | Intent-To-Treat |
| MCMC | Markov-Chain-Monte-Carlo |
| MMRM | Mixed Model Repeated Measures |
| NRS | Numeric Rating Scale |
| PCI | Potential Clinical Importance |
| PD | Pharmacodynamic |
| PDMP | Protocol Deviation Management Plan |
| PK | Pharmacokinetic |
| PRO | Patient reported Outcomes |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| TARC | Activation-regulated Chemokine |
| TA | Therapeutic Area |
| TFL | Tables, Figures & Listings |

### 12.8.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

### 12.9. Appendix 9: List of Data Displays

### 12.9.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|-------------------------------|-------------|------------|
| Study Population | 1.1 to 1.10 | N/A |
| Efficacy | 2.1 to 2.7 | N/A |
| Safety | 3.1 to 3.40 | 3.1 to 3.2 |
| Pharmacokinetic | 4.1 | 4.1 to 4.2 |
| Pharmacodynamic and Biomarker | 5.1 to 5.2 | 5.1 to 5.2 |
| Section | List | ings |
| ICH Listings | 1 to 26 | |
| Other Listings | 27 t | o 40 |

### 12.9.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required example mock-up displays provided in Appendix 10: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|-------------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Efficacy | EFF_Fn | EFF_Tn | EFF_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Pharmacodynamic and Biomarker | PD_Fn | PD_Tn | PD_Ln |

### NOTES:

Non-Standard displays are indicated in the 'IDSL / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.

### 12.9.3. Deliverables

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC | Final Statistical Analysis Complete |

### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort

# 12.9.4. Study Population Tables

| Study I | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL/ Example<br>Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1.1. | ITT | ES1 | Subject Status and Reason for Study Withdrawal | ICH E3, FDAAA, EudraCT | SAC |
| 1.2. | ITT | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | ICH E3 | SAC |
| 1.3. | Screened | ES6 | Summary of Screening Status and Reasons for Screen Failure | Journal Requirements Add Footnote "Note: Re-screened participants who have been randomised are included both in ENROLLED as well as FAILED category. | SAC |
| 1.4. | Enrolled | NS1 | Summary of Number of Participants Enrolled by Country and Site ID | EudraCT/Clinical Operations | SAC |
| Popula | tion Analysed | | | | |
| 1.5. | Screened | SP1 | Summary of Study Populations | IDSL | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 1.6. | ITT | DM1 | Summary of Demographic and Baseline Characteristics | ICH E3, FDAAA, EudraCT<br>Include: Baseline Eosinophil counts and<br>Fitzpatrick skin type | SAC |
| 1.7. | ITT | DM11 | Summary of Age Ranges | EudraCT Note: Include Age categories: Adult (18 – 64 years), >=65 – 84 years and >=85 years. | SAC |
| 1.8. | ITT | DM5 | Summary of Race and Racial Combinations | ICH E3, FDA, FDAAA, EudraCT | SAC |

| Study P | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. Population IDSL/ Example Shell Title Programming Notes Deliverable | | | | | |
| Prior ar | d Concomitan | t Medications | | | |
| 1.9. | ITT | MH1 | Summary of Past Medical Conditions | ICH E3 | SAC |
| Exposu | Exposure | | | | |
| 1.10. | 1.10. Safety POP_T1 Summary of Exposure to Study Treatment ICH E3 SAC | | | | |

# 12.9.5. Efficacy Tables

| Efficacy | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL/ Example<br>Shell | Title | Programming Notes | Deliverable |
| IGA | | | | | |
| 2.1. | ITT | EFF_T1 | Bayesian Posterior Probability for Comparison between Mepolizumab and Placebo | Note: Non-Responder imputation will be used | SAC |
| 2.2. | ITT | EFF_T2 | Number (%) of Participants in Each Category of the Investigator's Global Assessment Scale at Each Visit | | SAC |
| 2.3. | ITT | EFF_T3 | Summary of Proportion of Participants with IGA Score of 0 or 1 and at Least a 2-Grade Improvement from Baseline at Each Visit | Note: Non-Responder imputation will be used | SAC |
| EASI | | | | | |
| 2.4. | ITT | EFF_T4 | Summary of Change from Baseline/Percent Change from Baseline in EASI Score at Each Visit | Note: CFB, %CFB in bylines | SAC |
| 2.5. | ITT | EFF_T4 | Summary of Change from Baseline/Percent Change from Baseline in EASI Score at Each Visit by Baseline Blood Eosinophil Count Quartiles | Note: Include Quartiles categories as <=Q1(x), >Q1(x) - <=Q2, >Q2(x) - <=Q3(x) and >Q3(x). Include all quartiles value(x) | SAC |
| 2.6. | ITT | EFF_T5 | Summary of Proportion of Participants with >=50% and >=75% Improvement in EASI Score from Baseline at Each Visit | Note: >=50%, >=75% improvement in bylines. | SAC |
| Patien | Patient Reported Outcomes | | | | |
| 2.7. | ITT | EFF_T4 | Summary of Change from Baseline in Weekly Average of Daily Itch/pruritus NRS Score (based on Item #1 of Daily Sign and Symptom Severity Diary) at Each Visit | Includes Baseline values. Note: Mean change from baseline will be presented to only Week 4, 8, 12, 16 and 20 | SAC |

# 12.9.6. Safety Tables

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events (AEs) | | | | |
| 3.1. | Safety | AE1 | Summary of All On-Treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.2. | Safety | AE1 | Summary of All Post-Treatment Adverse Events by System Organ Class and Preferred Term | ICH E3 | SAC |
| 3.3. | Safety | AE15 | Summary of Common (>=3%) On-Treatment Non-Serious<br>Adverse Events by System Organ Class and Preferred Term<br>(Number of Participants and Occurrences) | FDAAA, EudraCT | SAC |
| 3.4. | Safety | AE1 | Summary of Adverse Events Reported on the Day of Dosing by System Organ Class and Preferred Term | | SAC |
| 3.5. | Safety | AE1 | Summary of On-Treatment Adverse Events by Highest Binding Antibody Result | | SAC |
| Serious | s and Other Sig | nificant Adverse l | -<br>Events | | · |
| 3.6. | Safety | AE16 | Summary of On-Treatment Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAA, EudraCT | SAC |
| 3.7. | Safety | AE16 | Summary of Post-Treatment Serious Adverse Events by System Organ Class and Preferred Term (Number of Participants and Occurrences) | FDAA, EudraCT | SAC |
| 3.8. | Safety | AE3 | Summary of Fatal Serious Adverse Events by Overall Frequency | | SAC |
| Advers | e Events of Sp | ecial Interest (AES | Sl's) | | |
| 3.9. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest<br>Reported by the Investigator as Meeting the Criteria for<br>Anaphylaxis | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.10. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis | Produced only if more than one AESI reported in this category. | SAC |
| 3.11. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest<br>Reported by the Investigator as Systemic Reactions - Allergic<br>(Type I Hypersensitivity) and Other Systemic | | SAC |
| 3.12. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) and Other Systemic | Produced only if more than one AESI reported in this category. | SAC |
| 3.13. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Reported by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | | SAC |
| 3.14. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Systemic Reactions - Allergic (Type I Hypersensitivity) | Produced only if more than one AESI reported in this category. | SAC |
| 3.15. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest<br>Reported by the Investigator as Systemic Reactions - Other<br>Systemic | | SAC |
| 3.16. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Systemic Reactions - Other Systemic | Produced only if more than one AESI reported in this category. | SAC |
| 3.17. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Reported by the Investigator as Local Injection Site Reactions | | SAC |
| 3.18. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Local Injection Site Reactions | Produced only if more than one AESI reported in this category. | SAC |
| 3.19. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Categorised as Serious Cardiac, Vascular and Thromboembolic Events | | SAC |

| Safety: | Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 3.20. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events of Special Interest Categorised as Serious Cardiac, Vascular and Thromboembolic Events | Produced only if more than one AESI reported in this category. | SAC |
| 3.21. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Categorised as Serious Ischemic Events | | SAC |
| 3.22. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events of Special Interest Categorised as Serious Ischemic Events | Produced only if more than one AESI reported in this category. | SAC |
| 3.23. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Categorised as Malignancies | | SAC |
| 3.24. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events of Special Interest Categorised as Malignancies | Produced only if more than one AESI reported in this category. | SAC |
| 3.25. | Safety | SAF_T1 | Summary of On-Treatment Adverse Events of Special Interest Categorised as Opportunistic Infections | | SAC |
| 3.26. | Safety | SAF_T2 | Summary Profile of On-Treatment Adverse Events of Special Interest Categorised as Opportunistic Infections | Produced only if more than one AESI reported in this category. | SAC |
| Labora | tory: Chemistry | y | | • | |
| 3.27. | Safety | LB1 | Summary of Chemistry Changes from Baseline | ICH E3<br>Includes Baseline values. | SAC |
| 3.28. | Safety | LB3 | Summary of Chemistry Shifts from Baseline Relative to Normal Range | | SAC |
| 3.29. | Safety | LB3 | Summary of Emergent Chemistry Results (Relative to the Potential Clinical Concern Range) | ICH E3 | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Labora | Laboratory: Haematology | | | | |
| 3.30. | Safety | LB1 | Summary of Haematology Changes from Baseline | ICH E3 Includes Baseline values. | SAC |
| 3.31. | Safety | LB3 | Summary of Haematology Shifts from Baseline Relative to Normal Range | | SAC |
| 3.32. | Safety | LB17 | Summary of Emergent Haematology Results (Relative to the Potential Clinical Concern Range) | ICH E3 | SAC |
| ECG | • | | | | |
| 3.33. | Safety | EG1 | Summary of ECG Findings | The ECG findings to be summarized are the ECG interpretation, clinical significance of abnormal ECGs | SAC |
| 3.34. | Safety | EG2 | Summary of Change from Baseline in ECG Values by Visit | Includes Baseline values. | SAC |
| 3.35. | Safety | EG10 | Summary of Actual and Change from Baseline QTc(F) Values by Category | Category column will be replaced and created based on the information provided in the Section 8.4.1. For Anytime Post-Baseline, the highest post-baseline QTcF value and the change from baseline for this highest post-baseline QTc value is categorised | SAC |
| Vital Si | gns | | | | |
| 3.36. | Safety | VS1 | Summary of Change from Baseline in Vital Signs | Includes Baseline values. | SAC |
| 3.37. | Safety | VS3 | Summary of Worst Case Vital Signs Results by PCI Criteria Post-Baseline Relative to Baseline | | SAC |

| Safety: | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Immun | genicity | | | | |
| 3.38. | Safety | SAF_T3 | Summary of Binding Antibody by Visit | | SAC |
| 3.39. | Safety | SAF_T4 | Summary of Neutralising Antibody by Visit | | SAC |
| 3.40. | Safety | SAF_T5 | Summary of Binding Antibody Assay Results: Highest Treatment<br>Emergent Confirmatory Result Any Time Post Baseline | | SAC |

# 12.9.7. Safety Figures

| Safety: | Safety: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Laborat | Laboratory | | | | |
| 3.1. | Safety | LIVER14 | Scatter Plot of Maximum vs. Baseline for ALT | IDSL Note: Figure created as no liver events report, but such a plot may flag participants who were not reported. | SAC |
| 3.2. | Safety | LIVER9 | Scatter Plot of Maximum ALT vs. Maximum Total Bilirubin | IDSL | SAC |

### 12.9.8. Pharmacokinetic Tables

| Pharmacokinetic: Tables | | | | |
|---|---|---|---|---|
| No. | No. Population IDSL / Example Shell Title Programming Notes | | | |
| 4.1. | PK | PKCT1 | Summary of Plasma Mepolizumab Pharmacokinetic Concentration-Time Data | SAC |

# 12.9.9. Pharmacokinetic Figures

| Pharmaco | Pharmacokinetic: Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| 4.1. | PK | PK_F1 | Scatter Plot of Individual Plasma Concentration Data by Participants' ADA Status | Note: Participants' ADA status is highest ADA result (Positive or Negative) in any post bassline visit. | SAC |
| 4.2. | PK | PK_F1 | Scatter Plot of Individual Plasma Concentration Data (with Mean $\pm$ SD) | Include Mean ± SD for each visit along with the individual plasma conc. data | SAC |

## 12.9.10. Pharmacodynamic and Biomarker Tables

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Blood E | Eosinophil Cou | nts | | | |
| 5.1. | Safety | PD_T1 | Summary of Blood Eosinophils Count at Each Visit | Include both absolute and ratio to baseline for log transformed blood eosinophil count. | SAC |
| 5.2. | Safety | PD_T2 | Summary of Mixed Model Repeated Measures (MMRM) Analysis for Blood Eosinophils Count | | SAC |

# 12.9.11. Pharmacodynamic and Biomarker Figures

| Pharma | Pharmacodynamic and Biomarker: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Blood E | osinophil Cou | nts | | | |
| 5.1. | Safety | PD_F1 | Scatter Plot of Individual Absolute Blood Eosinophils Count by Participants' ADA status | Note: Participants' ADA status is highest ADA result (Positive or Negative) in any post bassline visit. | SAC |
| 5.2. | Safety | PD_F2 | Plot of Least Squares Geometric Means and 95% CI of Ratio to Baseline in Blood Eosinophil Count | | SAC |

# **12.9.12. ICH Listings**

| ICH: Li | stings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Subjec | t Disposition | | | | |
| 1. | Screened | ES7 | Listing of Reasons for Screen Failure | Journal Guidelines | SAC |
| 2. | ITT | ES2 | Listing of Reasons for Study Withdrawal | ICH E3 | SAC |
| 3. | ITT | SD2 | Listing of Reasons for Study Treatment Discontinuation | ICH E3 | SAC |
| 4. | ITT | BL1 | Listing of Participants for Whom the Treatment Blind was Broken | ICH E3 | SAC |
| 5. | ITT | TA1 | Listing of Planned and Actual Treatments | IDSL | SAC |
| Protoc | ol Deviations | | | | |
| 6. | ITT | DV2 | Listing of Important Protocol Deviations | ICH E3 | SAC |
| 7. | ITT | IE3 | Listing of Participants with Inclusion/Exclusion Criteria Deviations | ICH E3 | SAC |
| Demog | raphic and Bas | eline Characteris | tics | | |
| 8. | ITT | DM2 | Listing of Demographic and Baseline Characteristics | ICH E3 Include Baseline Eosinophil Count and Fitzpatrick skin type | SAC |
| 9. | ITT | DM9 | Listing of Race | ICH E3 | SAC |
| Prior a | nd Concomitan | t Medications | | | |
| 10. | ITT | CM3 | Listing of Concomitant Medications | ICH E3 | SAC |
| Exposu | ıre | | | | |
| 11. | Safety | EX3 | Listing of Exposure Data | ICH E3 | SAC |

| ICH: Li | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Advers | e Events | | | | |
| 12. | Safety | AE8 | Listing of All Adverse Events | ICH E3 | SAC |
| 13. | Safety | AE7 | Listing of Participant Numbers for Individual Adverse Events | ICH E3 | SAC |
| 14. | Safety | AE2 | Listing of Relationship Between Adverse Event System Organ Classes, Preferred Terms, and Verbatim Text | IDSL | SAC |
| 15. | Safety | AE8 | Listing of Adverse Events Leading to Withdrawal from Study / Permanent Discontinuation of Study Treatment | | SAC |
| 16. | Safety | AE8 | Listing of Adverse Events Reported on the Day of Dosing | | SAC |
| 17. | Safety | AE8 | Listing of All Adverse Events of Special Interest | Produced only if more than one AESI reported. | |
| All Lab | oratory | | | | |
| 18. | Safety | LB5 | Listing of All Chemistry Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 19. | Safety | LB5 | Listing of All Haematology Laboratory Data for Participants with Any Value of Potential Clinical Importance | ICH E3 | SAC |
| 20. | Safety | LB14 | Listing of Laboratory Data with Character Results | | SAC |
| 21. | Safety | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | |
| 22. | Safety | LIVER13 | Listing of Subjects Meeting Hepatobiliary Laboratory Criteria Post-Baseline | | |
| ECG | • | | | <u> </u> | <u>.</u> |
| 23. | Safety | EG3 | Listing of ECG Values (Participants with QTcF >500 msec or Increase > 60 msec from Baseline) | | SAC |
| 24. | Safety | EG5 | Listing of Abnormal ECG Findings | IDSL | SAC |

| ICH: Lis | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable |
| Vital Si | gns | | | | |
| 25. | Safety | VS4 | Listing of All Vital Signs Data for Participants with Any Value of Potential Clinical Importance | IDSL | SAC |
| Immun | ogenicity | | | | |
| 26. | Safety | IMM2 | Listing of Immunogenicity Results | IDSL. Include columns for Screening<br>Binding Assay, Confirmation Antibody<br>Assay, Confirmation Assay Titre,<br>Transient/Persistent, Neutralizing<br>Antibody Assay | SAC |

# 12.9.13. Non-ICH Listings

| Non-IC | H: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| IGA | | | | | |
| 27. | ITT | EFF_L1 | Listing of Investigator's Global Assessment (IGA) Score | Note: Include Character result, Numeric score & CFB | SAC |
| EASI ar | nd %BSA | | | | |
| 28. | ITT | EFF_L2 | Listing of Eczema Area and Severity Index (EASI) Score | Note: Include Character result, Numeric score, CFB & %CFB | SAC |
| 29. | ITT | EFF_L4 | Listing of Total Body Surface Area (%BSA) | Note: Include Numeric score & CFB | SAC |
| Patient | -Reported Outo | comes | | | |
| 30. | ITT | EFF_L3 | Listing of Weekly Average of Daily itch/ pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary) | Note: Include Numeric score & CFB for all derived visits | SAC |
| 31. | ITT | EFF_L4 | Listing of Daily Sign and Symptom Severity Diary | Note: Include Numeric score | SAC |
| 32. | ITT | EFF_L4 | Listing of Patient Global Impression of Change Scores | Note: Severity of eczema symptoms and Severity of itch in by-lines. Note: Include Character result, Numeric score | SAC |
| 33. | ITT | EFF_L4 | Listing of Patient Global Impression of Severity Scores | Note: Include Character result, Numeric score & CFB | SAC |
| 34. | ITT | EFF_L4 | Listing of Clinician Global Impression of Change Scores | Note: Include Character result, Numeric score | SAC |
| PK | | | | | |
| 35. | PK | PKCL1P | Listing of Plasma Mepolizumab Concentration Time Data | | SAC |

| Non-ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Blood E | osinophil Cou | nts and Biomarke | rs | | |
| 36. | Safety | EFF_L4 | Listing of Blood Eosinophil Counts | Include both absolute and ratio to baseline blood eosinophil count | |
| 37. | Safety | N/A | Listing of Raw SAS Output for Mixed Model Repeated Measures (MMRM) Analysis for Blood Eosinophils Count | | |
| 38. | PD | EFF_L4 | Listing of Serum Free and Total Serum IL-5 Levels | | |
| 39. | PD | EFF_L4 | Listing of Serum Biomarker Endpoints | | |
| 40. | ITT | N/A | Listing of Raw SAS output of Bayesian Analysis of Response Rate in Investigator's Global Assessment (IGA) Score | | |

## 12.10. Appendix 10: Example Mock Shells for Data Displays

Example: POP T1 Page 1 of n

Protocol: 205050 Population: Safety

Table 1.10 Summary of Exposure to Study Treatment

| | | Placebo SC (N=xx) | Mepolizumab 100mg SC (N=xx) |
|---|---|---|---|
| Treatments Administered | n | 68 | 68 |
| | Mean | 11.6 | 12.7 |
| | SD | 3.30 | 1.33 |
| | Median | 13.0 | 13.0 |
| | Min. | 2 | 4 |
| | Max. | 14 | 14 |
| Number of Treatments | 1 | 0 | 0 |
| | 2 | 2 (3%) | 0 |
| | 3 | 3 (4%) | 0 |
| | 4 | 3 (4%) | 1 (1%) |
| Number of Days on Treatment | n | 68 | 68 |
| Number of bays on freatment | Mean | 330.8 | 357.2 |
| | SD | 91.43 | 37.39 |
| | Median | 365.0 | 365.0 |
| | Min. | 57 | 114 |
| | Max. | 394 | 392 |

205050

Note: Number of Days on Treatment = (Treatment Stop Date - Treatment Start Date) + another 28 days inclusive.

205050

Example: EFF\_T1 
Protocol: 205050

Population: Intent-to-Treat

Table 2.1
Bayesian Posterior Probability for Comparison between Mepolizumab and Placebo

| Visit | Treatment | n | Posterior<br>Mean<br>Response<br>Rate (80%<br>Cred Int) | Posterior<br>Median<br>Response Rate<br>(80% Cred Int) | Posterior<br>Mean<br>Difference<br>(80% Cred<br>Int) | Posterior<br>Probability<br>of Response<br>Rate ≥ 40% | - |
|---|---|---|---|---|---|---|---|
| Week<br>16 | Mepolizumab<br>100 mg SC | XX | xx.xx<br>(xx.xx,<br>xx.xx) | xx.xx<br>(xx.xx, xx.xx) | xx.xx<br>(xx.xx,<br>xx.xx) | xx.xx | xx.xx |
| | Placebo SC | XX | xx.x x<br>(xx.xx,<br>xx.xx) | xx.xx<br>(xx.xx, xx.xx) | | | |

Note: A Responder is defined as a subject who has an IGA score of 0 or 1 and a minimum 2-grade improvement from baseline. If a subject withdraws early from the study the due to lack of efficacy or disease progression, then all weeks after withdrawal they are assigned to be a non-responder.

Note: 0=Clear; 1=Almost Clear; 2=Mild; 3=Moderate; 4=Severe.

205050

Example: EFF\_T2

Protocol: 205050 

Population: Intent-to-Treat

Table 2.2

Number (%) of Subjects in Each Category of the Investigator's Global Assessment Scale at Each Visit

| Visit | Category | Placebo SC (N=XX) | Mepolizumab 100 mg SC (N=XX) |
|-------|--------------|-------------------|------------------------------|
| Day 1 | | (10 2222) | (14 2222) |
| | n | XX | XX |
| | Clear | XX (XX%) | XX (XX%) |
| | Almost Clear | XX (XX%) | XX (XX%) |
| | Mild | XX (XX%) | XX (XX%) |
| | Moderate | XX (XX%) | XX (XX%) |
| | Severe | XX (XX%) | XX (XX%) |

Programming note: Repeat for all study visits

205050

Example: EFF\_T3

Protocol: 205050

Protocol: 205050 

Population: Intent-to-Treat

Table 2.3

Summary of Proportion of Subjects with an IGA Score of 0 or 1 and at Least a 2-Grade Improvement from Baseline at Each Visit

| Visit | IGA score of 0 or<br>1 and at least a<br>2-grade<br>improvement | Placebo SC (N=XX) | Mepolizumab<br>100mg SC<br>(N=XX) | Proportions<br>Difference | 90% CI for<br>the<br>Proportions<br>Difference |
|---|---|---|---|---|---|
| Week 4 | n<br>Yes | XX (XX%) | XX<br>XX (XX%) | XX% | (XX.X%, |
| | No | XX (XX%) | XX (XX%) | | XX.X%) |

Note: A Responder is defined as a subject who has an IGA score of 0 or 1 and a minimum 2-grade improvement from baseline. If a subject withdraws early from the study the due to lack of efficacy or disease progression, then all weeks after withdrawal they are assigned to be a non-responder.

Note: Day 1 is considered as baseline.

Note: 0=Clear; 1=Almost Clear; 2=Mild; 3=Moderate; 4=Severe.

Programming note: Repeat for all available visits

205050

Example: EFF\_T4

Protocol: 205050 

Population: Intent-to-Treat

Table 2.4

Summary of Change from Baseline/Percent Change from Baseline in EASI Score at Each Visit

| Change from Baseline | | |
|---|---|---|
| | Placebo SC | Mepolizumab 100mg SC |
| | (N=XX) | (N=XX) |
| n | XX | XX |
| Mean | X • X | X.X |
| SD | X.XX | X.XX |
| Median | X • X | X.X |
| Min. | X | X |
| Max. | Χ | X |
| n | XX | XX |
| Mean | X • X | X.X |
| SD | X.XX | X.XX |
| Median | X • X | X.X |
| Min. | Χ | X |
| Max. | X | X |
| | Mean SD Median Min. Max. n Mean SD Median Min. | Placebo SC (N=XX) n XX Mean X.X SD X.XX Median X.X Min. X Max. X n XX Mean X.X Mean X.X Mean X.X Mean X.X Mean X.X Mean X.X Mean X.X Min. X Median X.X |

Summary: Percentage Change from Baseline

.....[Format as Change from Baseline]

Note: Day 1 is considered as baseline and summarized for absolute value. Programming note: Repeat for all available visits and include percent change from baseline

205050

Example: EFF\_T5

Protocol: 205050 

Population: Intent-to-Treat

Table 2.6

Summary of Proportion of Subjects with >=50% and >=75% Improvement in EASI Score from Baseline at Each Visit

| Visit | Improvement in EASI Score from | Placebo SC (N=XX) | Mepolizumab<br>100mg SC | Proportions<br>Difference | 90% CI for the Proportions |
|---|---|---|---|---|---|
| | baseline | | (N=XX) | | Difference |
| Week 4 | n | XX | XX | | |
| | >=50% improvement | XX (XX%) | XX (XX%) | XX% | (XX.X%, XX.X%) |
| | >=75% improvement | XX (XX%) | XX (XX%) | XX% | (XX.X%, XX.X%) |

205050

Example: SAF\_T1 Page 1 of n

Protocol: 205050

Population: Intent-to-Treat

Table 3.9

Summary of On-Treatment Adverse Events of Special Interest Reported by the Investigator as

| | g the Criteria for Anaphylaxi<br>Placebo SC<br>(N=XX) | Mepolizumab 100mg SC (N=XX) |
|---|---|---|
| Number of Subjects with Any Event | xx (xx%) | xx (xx%) |
| Hypersensitivity | | |
| Number of Subjects with Any Event<br>Facial Paralysis<br>Flushing<br>Injection related reaction<br>Rash | XX (XX%) XX (XX%) XX (XX%) XX (XX%) XX (XX%) | XX (XX%) XX (XX%) XX (XX%) XX (XX%) XX (XX%) |

### Other Systemic Reactions

| Number of Subjects with Any Event | XX | (XX%) | XX | (XX%) |
|-----------------------------------|----|-------|----|-------|
| Facial Paralysis | XX | (XX%) | XX | (XX%) |
| Flushing | XX | (XX%) | XX | (XX%) |
| Injection related reaction | XX | (XX%) | XX | (XX%) |
| Rash | XX | (XX%) | XX | (XX%) |

Example: SAF\_T2
Protocol: 205050

Protocol:  $20\overline{5}050$  Page 1 of n

Population: Safety

Table 3.10

Summary Profile of On-Treatment Adverse Events Reported by the Investigator as Meeting the Criteria for Anaphylaxis

| | Placebo<br>(N=xx) | Mepolizumab 100 mg SC (N=xx) |
|---|---|---|
| All Events<br>>=1 event [1] | 3/2 (3%) | 5/5 (7%) |
| <pre>1 event 2 events 3 events &gt;=4 events</pre> | 1 (1%)<br>1 (1%)<br>0 | 5 (7%)<br>0<br>0 |
| Serious Events<br>>=1 event [1] | 1/1 (1%) | 0 |
| <pre>Events considered related to Investigational Product &gt;=1 event [1]</pre> | 1/1 (1%) | 1/1 (1%) |
| Intensity [1] Mild Moderate Severe | 0<br>2/2 (3%)<br>1/1 (1%) | 4/4 (6%)<br>1/1 (1%)<br>0 |
| Outcome [1] Recovered/Resolved Recovering/Resolving Not Recovered/Not Resolved | 3/2 (3%)<br>0<br>0 | 5/5 (7%)<br>0<br>0 |

205050

| Recovered/Resolved With Sequelae | 0 | 0 |
|----------------------------------|----------|----------|
| Fatal | 0 | 0 |
| Action Taken [1] | | |
| Drug withdrawn | 0 | 0 |
| Dose reduced | 0 | 0 |
| Dose increased | 0 | 0 |
| Dose not changed | 3/2 (3%) | 5/5 (7%) |
| Dose interrupted | 0 | 0 |
| Not applicable | 0 | 0 |
| No. doses prior to event [1] | | |
| 1 | 0 | 0 |
| 2 | 0 | 1/1 (1%) |
| 3 | 0 | 0 |
| 4 | 0 | 1/1 (1%) |
| No. doses prior to first event | | |
| 1 | 0 | 0 |
| 2 | 0 | 1 (1%) |
| 3 | 0 | 0 |
| 4 | 0 | 1 (1%) |

<sup>[1]</sup> Information presented as number of events / number (%) participants with at least one event. Subjects may be counted in more than one row.


Example: SAF\_T3
Protocol: 205050
Population: Safety

Table 3.38 Summary of Binding Antibody by Visit

| Visit | Assay Result | | | Mepolizumab 100 mg SC (N=68) |
|---|---|---|---|---|
| Baseline | n<br>Negative<br>Positive | | xx<br>xx (xx%)<br>xx (xx%) | |
| | Titer Value | Median<br>Min.<br>Max. | 32.0<br>32<br>32 | 32.0<br>32<br>32 |
| Week 4 | n<br>Negative<br>Positive<br>Transient Po<br>Persistent Po | | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| | Titer Value | Median<br>Min.<br>Max. | 32.0<br>32<br>32 | 32.0<br>32<br>32 |
| Anytime Post Baseline | n<br>Negative<br>Positive<br>Transient Po | ositive | xx<br>xx (xx%)<br>xx (xx%) | xx (xx%) |

205050

| Persistent | Positive | xx (xx%) | xx (xx%) |
|-------------|----------|----------|----------|
| Titer Value | Median | 32.0 | 32.0 |
| | Min. | 32 | 32 |
| | Max. | 32 | 32 |

Note: The values shown at the anytime post baseline visit are based on each participants highest post baseline titer.

Any time post baseline would be Positive for a participants who had Negative and Positive post baseline results

205050

Example: SAF T4 Protocol: 205050

 Population: Safety

Table 3.39 Summary of Neutralising Antibody by Visit

| Visit | Assay<br>Result | Placebo<br>(N=xx) | Mepolizumab<br>100 mg SC<br>(N=xx) |
|---|---|---|---|
| Baseline | n<br>Negative<br>Positive | xx<br>xx (xx%)<br>xx (xx%) | xx (xx%) xx (xx%) |
| Week 4 | n<br>Negative<br>Positive | xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |
| Anytime Post Baseline | n<br>Negative<br>Positive | xx<br>xx (xx%)<br>xx (xx%) | xx (xx%)<br>xx (xx%) |

Note: NAb assay result only presented for participant with positive ADA assay. Any time post baseline would be Positive for a participant who had both Negative and Positive post baseline results.

205050

Example: SAF\_T5
Protocol: 205050

Protocol: 205050 

Population: Safety

Table 3.40

Summary of Binding Antibody Assay Results: Highest Treatment Emergent Confirmatory Result
Any Time Post Baseline

| Assay Result | Placebo<br>(N=xx) | Mepolizumab 100 mg SC (N=xx) |
|---|---|---|
| n<br>Negative<br>Positive<br>Transient Positive<br>Persistent Positive | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) | xx<br>xx (xx%)<br>xx (xx%)<br>xx (xx%)<br>xx (xx%) |
| Titer Value<br>Median<br>Min.<br>Max. | 32.0<br>32<br>32 | 32.0<br>32<br>32 |

Note: Includes only results from subjects who do not have a positive ADA assay prior to the first dose of investigational product.

205050

Example: PD\_T1
Protocol: 205050

Population: Intent-to-Treat

Table 5.1
Summary of Blood Eosinophil Count at Each Visit


| Visit | | , | 1 | | Mepolizumab<br>(N=68) | 100 mg SC |
|---|---|---|---|---|---|---|
| Baseline | Blood Eosinophils | (10^9/L) | n | <br>68 | 68 | |
| | | | Geo Mean | 0.172 | 0.177 | |
| | | | Std Logs | 1.3522 | 1.2890 | |
| | | | Median | 0.215 | 0.190 | |
| | | | Min. | 0.00 | 0.01 | |
| | | | Max. | 4.45 | 6.72 | |
| Week 4 | Blood Eosinophils | (10 <sup>9</sup> /L) | n | 66 | 66 | |
| | | | Geo Mean | 0.141 | 0.035 | |
| | | | Std Logs | 1.4972 | 0.9999 | |
| | | | Median | 0.195 | 0.040 | |
| | | | Min. | 0.00 | 0.00 | |
| | | | Max. | 3.35 | 1.56 | |
| | Blood Eosinophils F | Ratio to Baseline | n | 66 | 66 | |
| | - | | Geo Mean | 0.796 | 0.189 | |
| | | | Std Logs | 1.2976 | 1.1936 | |
| | | | Median | | 0.185 | |
| | | | Min. | 0.00 | 0.00 | |
| | | | Max. | 22.00 | 4.00 | |

Note: Data were log transformed.

Note: Where a result of zero was recorded, a small value (i.e. minimum all non-missing

results/2) was added prior to log transformation

205050

Example: PD\_T2


Population: Safety

Table 5.2

Summary of Mixed Model Repeated Measures (MMRM) Analysis for Blood Eosinophils Count

| Visit | Statistic | Placebo SC<br>N=xx | Mepolizumab 100 mg SC<br>N=xx |
|---|---|---|---|
| Week 4 | n | XX | XX |
| | LS Geometric Mean (SE) | x.xx (xx.xxx) | x.xx (xx.xxx) |
| | LS Geometric Mean Ratio to Baseline (SE) | x.xx (xx.xxx) | x.xx (xx.xxx) |
| | 95% Confidence Interval | (x.xx, x.xx) | (x.xx, x.xx) |
| | Treatment Ratio | | X.XX |
| | 95% Confidence Interval | | (x.xx, x.xx) |
| Week 8 | n | XX | XX |
| | LS Geometric Mean (SE) | x.xx (xx.xxx) | x.xx (xx.xxx) |
| | LS Geometric Mean Ratio to Baseline (SE) | x.xx(xx.xxx) | x.xx (xx.xxx) |
| | 95% Confidence Interval | (x.xx, x.xx) | (x.xx, x.xx) |
| | Treatment Ratio | | X.XX |
| | 95% Confidence Interval | | (x.xx, x.xx) |

Note: Treatment Ratio (Mepolizumab/Placebo) and 95% Confidence Intervals for Ratio to Placebo are obtained from MMRM model, with fixed categorical effects of Treatment, Visit, and Treatment-By-Visit Interaction and fixed continuous covariates of Baseline. 'XX' covariance structure was used.

Note: n is the number of participants with non-missing data at that visit.

205050

Example: EFF\_L1

Protocol:  $20\overline{5}050$  Page 1 of x

Population: Intent-to-Treat

Listing 24

Listing of Investigator's Global Assessment (IGA) Score

| Treatment | Site<br>ID./<br>Subj. | Visit/<br>Analysis<br>Visit | Date/<br>Study<br>Day | IGA<br>Character<br>result | IGA<br>Score | Change from Baseline score | Study<br>Treatment<br>Period | Follow-Up<br>Period | Relapsed (Y/N) |
|---|---|---|---|---|---|---|---|---|---|
| | XXX/<br>XXX | WEEK 2/ | | Moderate | | | | | |
| | XXX/<br>XXX | | | | | | | | |

<sup>[1]</sup> Participants who have an IGA score of 3 or 4 after achieving an IGA score of 0 or 1 and at least a 2-grade improvement during the Treatment and Follow-up Periods.

205050

Example: EFF\_L2
Protocol: 205050

Population: Intent-to-Treat


Listing 25

Listing of Eczema Area and Severity Index (EASI) Score

| Treatment | Site ID./<br>Subj. | Visit/<br>Analysis<br>Visit | Date/<br>Study<br>Day | EASI<br>Score | Change from<br>Baseline<br>Score | Study<br>Treatment<br>Period | Follow-Up<br>Period | Relapsed(Y/N) [1] |
|---|---|---|---|---|---|---|---|---|
| | XXX/<br>XXX | WEEK 2/ | | | | | | |
| | XXX/<br>XXX | | | | | | | |

[1]: Participants who have an increase in EASI score of  $\geq$ 25% from baseline during the Treatment and Follow-up Periods

205050

Example: EFF\_L3
Protocol: 205050


Population: Intent-to-Treat

Listing 27

Listing of Weekly Average of Daily Itch/pruritus NRS score (based on Item #1 of Daily Sign and Symptom Severity Diary)

| Treatment | | Visit/<br>Analysis Visit | Numeric<br>Score | Change from Baseline<br>Score |
|---|---|---|---|---|
| | XXX/<br>XXX | WEEK 2/ | | |
| | XXX/<br>XXX | | | |

205050

Example: EFF\_L4
Protocol: 205050


Population: Intent-to-Treat

Listing of xxxxxx

| Treatment | Site ID./<br>Subj. | Visit/<br>Analysis Visit<br>[optional] | Date/<br>Study<br>Day | Character result [optional] | Numeric<br>Score | Change<br>from<br>Baseline<br>[optional] |
|---|---|---|---|---|---|---|
| | XXX/<br>XXX | WEEK 2/ | | | | |
| | XXX/<br>XXX | | | | | |

Programming Note: Include optional columns as required.

205050

Example: PK\_F1/PD\_F1 Protocol: 205050

Population: Intent-to-Treat


Figure 4.1 Scatter plot of Individual Plasma Concentration Data by Participants' ADA Status



Time (unit)

205050

Example: PD\_F2


Population: Intent-to-Treat

Figure 5.2 Plot of Least Squares Geometric Means and 95% CI of Ratio to Baseline in Blood Eosinophil Count

